# The effectiveness of implementing a best practice primary health care model for low back pain (BetterBack®) compared to current routine care in the Swedish context: An internal pilot study informed protocol for an effectiveness-implementation hybrid type 2 trial

Allan Abbott<sup>1,2\*</sup>, Karin Schröder<sup>1</sup>, Paul Enthoven<sup>1</sup>, Per Nilsen<sup>3</sup>, Birgitta Öberg<sup>1</sup>
<sup>1</sup>Department of Medical and Health Sciences, Division of Physiotherapy, Faculty of Health Sciences, Linköping University, SE-58183 Linköping, Sweden.

<sup>2</sup> Faculty of Health Science and Medicine, Bond University, Gold Coast, Queensland, 4229, Australia.

Allan Abbott\* - <u>allan.abbott@liu.se</u> (TEL: 0046 13 282495); Karin Schröder - <u>karin.schroder@liu.se</u>; Paul Enthoven - <u>paul.enthoven@liu.se</u>; Per Nilsen - <u>per.nilsen@liu.se</u>; Birgitta Öberg - birgitta.öberg@liu.se;

#### **ABSTRACT**

Introduction: Low back pain (LBP) is a major health problem commonly requiring health care. In Sweden, there is a user pull for the development, implementation and evaluation of a best practice primary health care model for low back pain best practice model of primary care for LBP.

Aim: The overall aim is to investigate if and how the BetterBack© model of care for LBP implemented with a multi-facetted strategy is potentially more effective than current routine care in the Swedish primary health care context. The specific trial objectives are to: (A) To improve and understand the mechanisms underlying changes in Health Care Practitioner (HCP) confidence, attitudes and beliefs for providing primary health care for patients with LBP (B) Improve and understand the mechanisms underlying illness beliefs, self-care enablement, pain, disability and quality of life in patients with LBP; (C) Evaluate the implementation process and cost-effectiveness of the BetterBack© model of care for LBP in the Swedish primary health care context.

Methods: This study is an effectiveness-implementation hybrid type 2 trial. This involves a prospective cohort study investigating implementation on the HCP level and a patient blinded, pragmatic cluster randomized controlled trial with longitudinal follow up at 3, 6 and 12 months post baseline for effectiveness on the patient level. A superiority trial design framework will be used. A parallel process and economic analysis will also be performed. Patients will be allocated to routine care (control group) or the BetterBack© model of care (intervention group) according to the schedule of a dog leg design with 2 assessments in routine care. Short and long term HCP and patient level quantitative effectiveness outcomes will be compared between experimental conditions will be conducted as well as causal mediation analysis. Qualitative HCP and patient level experiences of the BetterBack© model of care will also be investigated.

**Dissemination:** The findings will be published in peer-reviewed journals and presented at national and international conferences. Further national dissemination and implementation in Sweden and associated national quality register data collection are potential future developments of the project.

Trial registration: ClinicalTrials.gov: NCT03147300

**Date and version identifier:** 30 Sept 2017, protocol version 2.

**Key words:** Low back pain, model of care, effectiveness, implementation.

Word count: 7421 words

<sup>&</sup>lt;sup>3</sup> Department of Medical and Health Sciences, Division of Community Medicine, Faculty of Health Sciences, Linköping University, SE-58183 Linköping, Sweden.

<sup>\*</sup>Corresponding author

#### Strengths and limitations of this study

- This is the first study of effectiveness and implementation of a best practice model of care in LBP primary care in Sweden.
- An international consensus framework has been used for the development, implementation and evaluation of the models of care.
- The main trial's a priori methodology has been informed and refined by an initial internal pilot phase.

#### **BACKGROUND**

Low back pain (LBP) is one of the most prevalent and burdensome problems for individuals and society in Sweden and worldwide [1,2]. LBP is often defined in terms of its localization, duration, severity, frequency, and interference on activities of daily living [3]. Most new episodes of LBP are self-limiting with only approximately 20% having persistent symptoms but a large majority experience pain recurrence [1]. The aetiology of LBP is often classified as specific or non-specific, based upon if a pathoanatomical cause can be identified through objective diagnostic assessment and confirmed by medical imaging [4]. The prevalence of LBP caused by specific pathology of serious nature such as malignancy, spinal fracture, infection, or cauda equine syndrome requiring secondary or tertiary health care has been reported to range between < 1%-4% in the primary health care setting [5,6]. Furthermore, nerve root problems associated with radiculopathy or spinal stenosis are thought to explain approximately 5%-15% of cases [7,8]. Medical imaging studies have highlighted that approximately 50% of younger adults and 90% of older adults have degenerative findings and large variations in lumbar spine morphology [9]. This is however evident in both symptomatic and asymptomatic individuals suggesting that low back pain is more typically a result of benign dysfunctional biological and psychological functions as well as social contextual factors influencing the pain experience.

In Sweden, the health care process for patients with LBP tends to be fragmented with many health care practitioners (HCP) giving conflicting information and providing interventions of varying effectiveness [10,11]. Our studies have shown that only a third of patients on sick leave for musculoskeletal disorders receive evidence-based rehabilitation interventions in primary care [10,11]. Furthermore our research has also demonstrated that there are still interventions that physiotherapists in primary care consider to be relevant in clinical practice despite the absence of evidence or consensus about the effects [12]. Our preliminary data suggests that when patients with LBP are referred to a specialist clinics, up to 48% have not received adequate evidence-based rehabilitation in primary care. The development of clinical practice guidelines aims to provide HCP with recommendations based on strength of available evidence as well as professional consensus for the intervention's risk and benefits for the patients. Such guidelines are lacking in Sweden but have recently been developed by the Danish Health and Medicines Authority and the English National Institute for Health and Care Excellence [13-15]. These national guidelines provide a thorough assessment of current evidence and can be used in Sweden to form the basis for locally adapted recommendations that are feasible to integrate in local health care setting.

Common to LBP, central recommendations from evidence based clinical guidelines for arthritis are also education and exercise therapy aimed at improving patient self-care. These principles have been packaged in well-known models of care describing how complex patient interventions can be delivered by clinicians. These model of care include "Better Management of Patients with Osteoarthritis (BOA)" in Sweden [16] and "Good Life with Osteoarthritis" in Denmark (GLA:D) [17]. Annual reports from BOA and GLA:D indicate an HCP acceptance through a broad national use of the models of care [18,19]. Furthermore, improvements in patient reported pain, physical function and decreased use of pain medication after receiving these models of care have been reported [18,19]. There is currently a paucity of evidence to determine if and how a similar best practice model of care for LBP could improve therapist and patient rated outcomes in the primary

treatment and secondary prevention of LBP.

Recently an international consensus has been reached proposing a framework for the development, implementation and evaluation of musculoskeletal models of care [20]. The theoretical underpinning is important in developing a model of care aimed at behavioural change to understand and explain the mechanisms of change [20]. Social-cognitve theories are widely used to predict and explain behaviour change. For example, the Theory of Planned Behaviour (TPB) [21] can be utilised to explain how intentions and volition of behaviour such as HCP use of a model of care can potentially be influenced by an intervention aiming to strengthen associations with attitudes, social norms and perceived behavioural control concerning the model. Furthermore, the Common Sense Model of self-regulation (CSM) [22] can been utilised to explain how behavioural change such as improved patient reported pain, physical function, self-care enablement and quality of life can potentially be influenced by an intervention aiming to strengthen associations with improved patient cognitive and emotional illness representations and comprehensibility through coping procedures [22].

It is important to apply knowledge from implementation science to achieve effective implementation of a best practice model of care in primary health care [23-26]. Implementation science is the scientific study of uptake of research findings and evidence-based practices into routine practice to improve the quality and effectiveness of health care and services [27]. Implementation strategies focus on determinants minimising barriers and maximising enablers that impact on the implementation and use of evidence-based practices. Recent implementation science studies investigating the uptake of national clinical guidelines for LBP in Denmark and the Netherlands have found multifaceted strategies to facilitate HCP behaviour change to be more cost-effective than single-faceted strategies [28,29].

There is therefore a clear rationale for evaluating the extent to which and how a best practice primary health care model for low back pain (BetterBack©) implemented with a multi-facetted strategy is potentially effective in the Swedish context. This article describes the BetterBack© trial internal pilot and protocol for the main trial. The protocol conforms to the SPIRIT guidelines [30].

#### **AIMS**

The overall aim is to investigate the effectiveness of the BetterBack model of care for LBP implemented with a multi-facetted strategy in a Swedish primary health care context. The specific trial objectives are to: (A) To improve and understand the mechanisms underlying changes in HCP confidence, attitudes and beliefs for providing primary health care for patients with LBP (B) Improve and understand the mechanisms underlying illness beliefs, self-care enablement, pain, disability and quality of life in patients with LBP; (C) Evaluate the implementation process and cost-effectiveness of the BetterBack model of care for LBP in the Swedish primary health care context.

#### **HYPOTHESIS**

- 1. HCP reported confidence, attitudes and beliefs for providing primary health care for LBP will show statistically significant improvement after a multifaceted implementation of the BetterBack© model of care compared to baseline before implementation. Intentional and volitional HCP rated determinants of implementation behaviour regarding the BetterBack© model of care will mediate improved confidence, attitudes and beliefs in a causal effects model.
- 2. The multifaceted implementation of the BetterBack© model of care will result in more statistically significant and greater clinically important improvement compared to current routine care for LBP regarding patient-reported measures for illness beliefs, self-care enablement, pain, disability and quality of life. Improvements in illness beliefs will mediate

- the effect on these outcomes.
- 3. A multifaceted implementation of the BetterBack☺ model of care compared to current routine care will result in fewer patients with persisting LBP, fewer requiring specialist care and more statistically significant incremental cost-effectiveness ratio (ICER) based on cost per EuroQoL-5 Dimension Questionnaire (EQ-5D) quality-adjusted life years (QALY) gained.

#### **METHODS**

#### Study design

World Health Organization Trial Registration Data Set is presented in table 1. This study is an effectiveness-implementation hybrid type 2 trial [31]. This involves a prospective cohort study design investigating implementation on the HCP level and a patient blinded, pragmatic cluster randomized controlled trial with longitudinal follow up at 3, 6 and 12 months post baseline for effectiveness on the patient level. A superiority trial design framework will be used. A parallel process and economic analysis will also be performed. This design was chosen because the multifaceted implementation of the BetterBack© model of care will be first targeted at changing HCP level behaviour who will then in turn implement behavioral change strategies on a patient level. Randomisation at the patient level is not possible due to potential carry-over effects of the HCP transitioning back and forth between providing routine care or the BetterBack© model of care for different patients. Instead, patients will be allocated to routine care (control group) or the BetterBack© model of care (intervention group) depending upon the clinics allocation. Patients will remain in their allocated group throughout the study.

The main study design is a dog leg with 2 assessments in routine care [32,33]. This involves the first cluster being assessed after the implementation of the BetterBack® model of care. The second cluster is assessed after a period of current routine care (control), and assessed again after the implementation of the BetterBack® model of care. The third cluster will receive current routine care (control) throughout the trial. The initial implementation of the BetterBack® model of care in cluster 1 allows for an internal pilot to determine the HCP acceptability of the intervention and trial within the first cluster [34,35]. A progression criteria for continuing to the main trial requires that HCP who have completed the BetterBack® education workshop rate on average a maximum of 2.5 out of 5 on the following determinant of implementation behaviour question: I expect that the application of BetterBack® model of care will be useful (1 = agree completely - 5 = do not agree at all).

The internal pilot also monitors patient recruitment during the first 2 months to provide a check point to optimize the main study design while data generated will still contribute to the final analyses to maintain trial efficiency [34,35]. Clusters are expected to recruit and gather data for at least 20 LBP patients per month in the internal pilot. In the dogleg design it is possible to vary the time point of cluster 2 to cross forward from the control to intervention condition if the patient recruitment process in either cluster 1 or 3 is more or less than expected in the internal pilot. In the event that cluster 1 recruit less than expected and clusters 2 or 3 recruit more than expected, then cluster 2 will cross forward to the intervention condition immediately after the internal pilot. If cluster 1 recruit more than expected and cluster 2 or 3 recruit less than expected during the internal pilot phase, then cluster 2 will cross forward to the intervention condition later in the main trial to allow adequate current routine care data collection. Implementation of the BetterBack<sup>®</sup> model of care in cluster 3 will occur directly after the end of patient recruitment in cluster 3. The study design is outlined in table 2.

#### **Study setting**

The Östergötland public health care region has a total population of 453 596 inhabitants with approximately 5000 patients per year accessing primary care physiotherapy due to LBP. In the

public health care region of Östergötland, a large majority of consultations for LBP are via direct access to the 15 primary care physiotherapy rehabilitation clinics. A smaller percentage of consultations are via referral to these rehabilitation clinics from the 36 primary health care general practices in the region. Therefore the focus of this study is on the physiotherapeutic rehabilitation process for LBP in primary care. The rehabilitation clinics form three clusters in Östergötland health care region. These clusters are based on municipal geographical area and organisational structure of the rehabilitation clinics which helps to minimize contamination between separate clusters of clinics (Figure 1). Cluster west is comprised of 5 clinics with 27 physiotherapists, cluster central is comprised of 6 clinics with 44 physiotherapists and cluster east is comprised of 6 clinics with 41 physiotherapists.

#### Eligibility criteria

Registered physiotherapists practicing in the allocated clinics and regularly working with patients with LBP will be included in the study. These physiotherapists will assess the eligibility of consecutive patients before and after the implementation of the BetterBack<sup>®</sup> model of care based on the following criteria:

*Inclusion criteria:* Males and females 18-65 years; Fluent in Swedish; Accessing public primary care due to a current episode of a first-time or recurrent debut of benign low back pain with or without radiculopathy.

*Exclusion criteria:* Current diagnosis of malignancy, spinal fracture, infection, cauda equine syndrome, ankylosing spondylitis or systemic rheumatic disease, previous malignancy during the past 5 years; Spinal surgery during the last 2 years; Current pregnancy or previous pregnancy up to 3 months before consideration of inclusion; Patients that fulfil criteria for multimodal/multiprofessional rehabilitation for complex longstanding pain; Severe psychiatric diagnosis.

A signed patient consent form will be collected by the physiotherapist before baseline measures are collected and intervention is commenced according to the study protocol. The therapist's intervention will not be effected by the patient's decision to participate or not participate in the study, only data collected will not be performed for those not participating.

#### Interventions

#### Control condition – current routine physiotherapeutic care for LBP in primary health care

Patients attending rehabilitation clinic clusters that have not have not yet completed the implementation of the BetterBack© model of care will receive treatment as usual according to current routine care clinical pathways (Figure 2). A clinical pathway specified in Östergötland public health care region requires that for patients accessing primary care due to LBP, a triage is to be performed by licensed HCPs (Physiotherapists, Nurses or General Practitioners (GP)), to triage for specific pathology of serious nature. These approximately 1-4% of patients with suspected specific pathology of serious nature are then to be examined by GPs and referred for specific intervention in secondary or tertiary health care. The majority of patients with LBP who on initial triage are assessed as having benign first-time or recurrent debut of LBP are then scheduled for physiotherapy consultation and implementation of a LBP management plan. If the patient has persistent functional impairment and activity limitation despite 2-3 months of primary care intervention, the clinical pathway specifies inclusion criteria for specialist care referral pathways (Figure 2).

#### Intervention condition – The BetterBack@model of care for LBP

Development and design of the BetterBack@model of care for LBP

A framework for the development of musculoskeletal models of care [20] was used to guide

development of the BetterBack® model of care for LBP. The high prevalence and burden of LBP [1,2], discordance in evidence based rehabilitation processes [10-12], a lack of physiotherapeutic clinical practice guidelines and a user-pull for a best practice model of care requested by physiotherapy clinic managers in the Östergötland health care region have been identified in the primary care of LBP. Therefore, a case for change has been justified to improve current physiotherapeutic health service delivery for the primary care of LBP. The structure and components of BetterBack® where developed by engaging a work group of physiotherapy clinicians (clinical champions) from each primary care cluster in the Östergötland public health care region and physiotherapy academics at Linköping University. To identify which key areas of contemporary care were of relevance for BetterBack®, the following tasks were performed by the work group:

- 1) Discussion and outline of the current routine care clinical pathway for LBP and areas needing improvement: The work group concluded that a best practice model of care needed to focus on the primary care physiotherapy process outlined by the red square in figure 2.
- 2) Analysis and discussion of existing international evidence based guidelines: The following thorough and up-to-date systematic critical literature reviews and international clinical guidelines [13-15, 36] were analysed and discussed by the work group.
- 3) Adaptation of evidence based recommendations to the Swedish context: The development of evidence based recommendations was based the Swedish National Board of Health and Welfare methods for guideline construction [37]. The overall grade of evidence together with a consensus position based on professional experience and patient net benefit versus harms and costs are the key aspects on which the work group has formulated local recommendations to reflect their strength [38]. The recommendations have been externally reviewed by local spinal physicians and international experts from the University of Southern Denmark. A summary of the Östergötland health care region physiotherapeutic clinical practice guideline recommendations for primary care management of LBP with or without radiculopathy as well as the implementation tools used in the BetterBack© model of care is provided in the supplementary material to this protocol article.
- 4) Considering potential barriers to the uptake of evidence based recommendations by health care professionals [39] and patient adherence to LBP management interventions [40], the work group identified and discussed targeted physiotherapist and patient behaviour change priorities of relevance for BetterBack. The Behaviour Change Wheel [41] (figure 3) was used to describe how the BetterBack<sup>©</sup> model of care at the guideline policy level applies theory-informed HCP and patient focused intervention functions with specific behavioural change techniques [42]. To help understand the mechanism of action of behavioural change interventions, the Theoretical Domains Framework (TDF) [43] has been integrated into the Behavioural Change Wheel [41]. The TDF is comprised of 14 theoretical domains/determinants of behavioural change which can be matched with behavioural change techniques to understand their effect on the central source of behaviour [44]. The central source of behaviour in the behavioural change wheel is described by the COM-B model. In the COM-B model, a person's capability (physical and psychological), opportunity (social and physical) can influence on motivation (automatic and reflective) enacting behaviours that can then alter capability, motivation and opportunity [41]. The COM-B provides a broad model of behaviour where our causal assumptions of the BetterBack@ model of care which are adapted from the TPB on a HCP level [21] and also adapted from the CSM on a patient level [22] can be applied in the Behavioural Change Wheel [41].

The first step in the BetterBack© model of care is to target HCP behaviour for the adoption of the BetterBack© model of care. Impeding barrier behaviours requiring change include low awareness of the model, beliefs of negative consequences, a biomedical treatment orientation rather than a

biopsychosocial orientation and primarily low beliefs about skills/capabilities for improving self-care patient management. Once HCP behaviour change has occurred, this can influence behaviour change on a patient level targeting patient understanding of the mechanisms and natural course of benign LBP and patient enablement of self-care. Impeding barrier behaviours requiring change include maladaptive beliefs on the cause and persistent course of LBP (low outcome expectation, anxiety, catastrophizing, fear-avoidance, and negative illness beliefs), contextual factors, low self-care enablement and low baseline physical activity. The potential outcomes of behavioural change could be improved illness beliefs, self-care enablement, pain, function, quality of life and health care utilization. The specific BetterBack© intervention content and mechanism of action for HCP behavioural change is outlined in table 3. A flow-diagram describing the BetterBack© model of care patient intervention process is displayed in figure 4.

Multifaceted implementation strategy for the BetterBack@model of care

The multifaceted implementation strategy is composed of the following 3 main facets:

1) Forming an **implementation forum** including head of departments/managers of the rehabilitation units and the clinical researchers.

- The implementation forum will collaborate on deciding overarching goals, timeline and logistics facilitating the implementation of the BetterBack® model of care in primary care rehabilitation clinic clusters in the Östergötland public health care region.
- 2) Forming a **support team** comprised of experience clinicians as local supervisors and faculty researchers as knowledge facilitators.
  - The support team is composed by trusted clinicians with special skills in LBP treatment from each participating unit and have had involvement in the work group for local adaptation of the BetterBack© model of care in their health care region.
- 3) Forming a **package of education and training** that the support team can utilize to assist the use of the BetterBack© model of care by HCP.
  - Physiotherapists in the 3 geographical clusters of public primary care rehabilitation clinics in Östergötland will be offered to participate in a 13.5 hours (2 days), continued medical education (CME) workshop. The workshop is designed by the support team with at least 2 clinical researcher and 1 experienced clinician (clinical champion) from the rehabilitation unit cluster present in the support team's delivery of the workshop for each cluster. The HCP education provided in the workshop format is described in supplementary file 2.
  - Key components of the educational program are:
    - Education about evidence based recommendations for LBP care and the BetterBack© model of care through an experiential learning process applying problem based case studies and clinical reasoning tools.
    - Practical use of the standardized BetterBack© education and exercise programs aiming at self-care as well as function and activity restoration.
    - Access to a website describing the BetterBack model of care. A chat forum will give an opportunity for clinicians to ask questions and share different experiences of the new strategy managed by the support team. Researchers will respond to questions from the participating clinicians.
  - To consolidate education at the local clinics, the local support team member (clinical champion) will provide continued maintenance of education according to the BetterBack model.

#### **Outcomes**

#### HCP outcomes:

1. Primary outcome measure

• Practitioner Confidence Scale (PCS) [45] mean change from baseline to 3 months post baseline. Practitioner reported confidence is the primary HCP behavioural change goal for the HCP education and training workshop in the multifaceted implementation of the BetterBack© model of care. The 3 month time frame allows for the development and consolidation of HCP behavioural change after application in repeated patient cases.

#### 2. Secondary outcome measures

- PCS [45] mean immediate change from baseline to directly after the HCP education and training workshop as well as mean long term change from baseline to 12 months post baseline. This secondary outcome is important for the understanding of longitudinal HCP behavioural change.
- Pain Attitudes and Beliefs Scale for physical therapists (PABS-PT) [46] mean change from baseline, to directly after the HCP education and training workshop as well as at 3 and 12 months post baseline.

#### Patient outcomes:

#### 1. Primary outcome measure

- Numeric rating scale for lower back related pain intensity during the latest week (NRS-LBP) [47]. The mean difference between control and intervention groups in change between baseline and 3 months post baseline will be analysed. Pain intensity is the primary functional impairment that patients with LBP contact primary health care for and has been recommended by international consensus to be included as a core outcome domain for clinical trials in non-specific low back pain [48]. International consensus even recommends patient reported NRS change over 6 months as a core metric for pain management interventions [49].
- Oswestry disability index version 2.1(ODI) [50]. The mean difference between control and intervention groups in change between baseline and 6 months post baseline will be analysed. Disability, analogues to decreased physical functioning and activity limitation has been recommended by international consensus to be included as a core outcome domain for clinical trials in non-specific low back pain [48]. International consensus even recommends patient reported ODI change over 6 months as a core metric for functional restoration [49].

#### 2. Secondary outcome measures

- NRS-LBP [47] and ODI [50] mean difference between control and intervention groups in short-term change from baseline to 3 months post baseline and mean long-term change from baseline to 12 months post baseline. These secondary outcomes are important for the understanding of longitudinal patient-rated changes in pain intensity and disability after primary care intervention.
- The European Quality of Life Questionnaire (EQ-5D) [51]. The mean difference between control and intervention groups in change between baseline and 3, 6 and 12 months post baseline will be analysed. Health related quality of life has been recommended by international consensus to be included as a core outcome domain for clinical trials in non-specific low back pain [48]. International consensus even recommends patient reported EQ-5D change over 6 months as a core metric for pain management interventions [49].
- The Brief Illness Perception Questionnaire (BIPQ) [52]. The mean difference between control and intervention groups in change between baseline and 3, 6 and 12 months post baseline will be analysed. Illness perception has been shown to predict longitudinal pain and disability outcomes in several LBP studies [53-57].
- Patient Enablement Index (PEI) [58], Patient Global Rating of Change (PGIC) [59] and Patient Satisfaction (PS) [60] mean difference between control and intervention groups at 3, 6 and 12 months post baseline will be analysed.

#### Health care process outcomes:

#### 1. Primary outcome measure

• Proportional difference between control and intervention groups for incidence of

participating patients receiving specialist care for LBP between baseline and 12 months after baseline. Incidence proportion, analogous to cumulative incidence or risk is calculated by taking the number of patients receiving specialist care of LBP and dividing it by the total number of patients recruited to the study. The main goal of both the control and interventions conditions in primary care for benign first-time or recurrent debut of LBP is to improve patient reported outcomes without the need of secondary or tertiary health care processes.

#### 2) Secondary outcomes measures

- Mean difference between control and intervention groups for change between baseline and final clinical visit regarding grade of patient functional impairment and activity limitation according to the ICF brief core set for LBP [61].
- The proportion of patients who receive the BetterBack@ model of care.

#### Participant timeline

The trial timeline is shown in table 2. The intervention schedule started with the development of evidence based recommendations and the BetterBack© model of care which occurred during June 2016 - February 2017. The enrolment schedule started with cluster enrolment and randomisation in March 2017. This resulted in the first allocated cluster 1 (west) entering internal pilot of implementing the BetterBack© model of care HCP education and training workshop which occurred in March 2017. This was followed up with a 2 month internal pilot of patient enrolment schedule occurring in all 3 clusters during April-May 2017. In order to finalise a sample size calculation for the main trial, baseline data collected during the internal pilot is compared to follow-up data 3 months after baseline for the primary outcome measure questionnaires to analyse initial HCP and patient effects of the implementation of BetterBack© model of care in cluster 1 compared to the control conditions in clusters 2 & 3. In the transition to the main trial, patient enrolment and baseline assessments will then continue to occur until January 2018. The eventual time of crossing forward of cluster 2 into the implementation of the BetterBack© model of care is determined by the internal pilot trial results. Participants in the trial will be follow-up longitudinally at 3, 6 and 12 months after baseline measures. The schedule for assessments is also outlined in table 2.

#### Sample size

An initial sample size estimation in the planning stage of the study assumed at least a small Cohens d effect size (d=0.35) for the HCP behavioural change primary and secondary outcomes. This is based on previous literature showing small-moderate HCP behavioural change effects sizes using similar interventions to increase the uptake of evidence-based management of LBP in primary care [62-63]. Considering also a 1-tailed p = 0.05 for the benefit of the multifaceted implementation of BetterBack, 80% statistical power and a 20% loss to follow-up, a sample size of n = 63 HCP is needed for a matched pairs t-test statistics comparing baseline and follow-up means. We assume a possible carry-over of a similar effect size (d=0.35) on patient behavioural change primary and secondary outcomes. Considering also a 1-tailed p = 0.05 for the benefit of the multifaceted implementation of BetterBack© compared to usual care and a 80% statistical power, the number of patients required for an individually randomized simple parallel group design would be n = 204. Adjusting for the design effect due to clustering randomizing, an intracluster correlation of 0.01 and a cluster autocorrelation of 0.80, a dog leg design with 2 assessments in routine care and 100 patients in each cluster section would require at least n = 402 patients over 2.41 clusters according to algorithms described by Hooper & Bourke [32]. In a balanced recruitment schedule, this equates to 14 patient per months per cluster for a total of 3 clusters. Allowing for potential unbalanced recruitment flow and a potential drop-out in the longitudinal outcomes at 3, 6 and 12 months post baseline, each cluster will aim for up to 20 patients per month equating to a potential total study n = 600.

#### Recruitment

In an effort to curb recruitment difficulties, strategies to promote adequate enrolment of participants into the study will be used. We anticipate less problems with recruitment into the prospective cohort study design investigating the multifaceted implementation of the BetterBack@ model of care on the HCP level. This is due to the study having a user-pull endorsed by clinical department managers calling all HCP working with patients with LBP at their clinics to participate. However, recruitment of patients into the cluster randomized controlled trial is dependent upon the feasibility of recruitment processes adapted to the context of each individual clinic and the compliance of HCP to administer recruitment of consecutive patients. A strategy to optimise the administration of patient recruitment will involve the author KS regularly visiting participating clinics to inform HCP of the study protocol and help streamline practical administration of the protocol in the context of the individual clinics. KS will also monitor weekly recruitment rates from the clinics and provide motivational feedback on recruitment flow to clinical department managers and designated clinical champions who will provide additional motivational feedback to HCP. In accordance with a Consolidated Standards of Reporting Trials, a flow diagram displaying participant enrolment, allocation, follow-up and analysis will be constructed [64]. Reasons for exclusion, declined participation, protocol violations and loss to follow-up will be monitored by KS.

#### Allocation and blinding

Random concealed allocation of clusters was performed by a blinded researcher randomly selecting from 3 sequentially numbered, opaque, sealed envelopes. The method resulted in the following order: 1=cluster west, 2=cluster central and 3=cluster east. The author KS informed the clinics in the different clusters of their allocation to the control or intervention study condition. Due to the nature of the study and intervention, HCP conducting patient measurements and treatment cannot be blinded to group allocation. Risk of bias is minimal as the primary and secondary outcomes are patient self-reported questionnaires. Patients will be blinded to group allocation. The researcher responsible for statistical analysis will not be blinded to group allocation.

#### **Data collection**

#### HCP reported professional behaviour questionnaires:

- The PCS contains 4 items reported on 5-point Likert scales where a total score of 4 represents greatest self-confidence and 20 represents lowest self-confidence for managing patients with LBP. The structural validity in terms of internal consistency of the items have been shown to be good with a Cronbach α coefficient = 0.73 in a single factor model for self-confidence [45]. The questionnaire has been forward translated by our research group from English to Swedish.
- The PABS-PT consists of two factors where higher scores represent more treatment orientation regarding that factor. One factor with 10 items measures the biomedical treatment orientation (Score 0-60) and one with 9 items measures the biopsychosocial treatment orientation (Score 0-54) [45]. Each item is rated on a 6-point Likert scale ranging from 1='totally disagree' to 6='totally agree'. The internal consistency of the biomedical factor has been shown to be good with a range between Cronbach α=0.77-0.84. Futhermore, the biopsychosocial factor has been shown to be adequate with a range between Cronbach α=0.62-0.68 [65]. Construct validity and responsiveness to educational interventions has been shown to be positive along with the test-retest reliability with reported intra-class correlation coefficient (ICC) on the biomedical factor=0.81 and on the biopsychosocial factor=0.65 [65]. The questionnaire has been forward translated from English to Swedish in a previously published study [66].
- The Determinants of Implementation Behaviour Questionnaire (DIBQ) was originally constructed based on the domains of the TDF [43, 67]. Confirmatory factor analysis resulted in a modified 93 item questionnaire assessing 18 domains with sufficient discriminant validity. Internal consistency of the items for the 18 domains was good, ranging from 0.68-0.93 for the Cronbach α coefficient [68]. The questionnaire has been forward translated by

our research group from English to Swedish. After face validity consensus in our research group regarding relevant domains for the implementation of BetterBack© model of care, the questionnaire was shortened to the following domains: Knowledge, Skills, Beliefs about capabilities, Beliefs about consequences, Intentions, Innovation, Organisation, Patient, Social influence, Behavioural regulation totalling to 57 items. Questions were adapted to the context of HCP reported determinants of an "expected" implementation of BetterBack© model of care for measurement directly after the HCP education and training workshop. HCP reported determinants retained orginal wording for the questionnaires at 3 and 12 months after the implementation of BetterBack© model of care. The response scale used for each DIBQ question in our study is a 5-point Liket scale ranging from 1= 'totally agree' to 5='totally disagree'.

#### Patient reported outcome measures:

- NRS-LBP intensity during the latest week is an 11-point scale consisting of integers from 0 through 10; 0 representing "No pain" and 10 representing "Worst imaginable pain". Previous research in a LBP cohort has shown a test-retest reliability ICC = 0.61, a common standard deviation=1.64 points, the standard error of measure = 1.02 and minimal clinically important difference (MCID) in LBP after treatment=2 [69,70].
- ODI version 2.1 assesses patient's current LBP related limitation in performing activities such as personal care, lifting, walking, sitting, standing, sleeping, sex life, social life and travelling. The ODI consists of 10 items with response scales from 0 to 5, where higher values represent greater disability. The ODI is analysed as a 0 to 100 percentage variable where lower scores represent lower levels of low back pain disability. A reduction of 10 points is considered the MCID in LBP after treatment [50,70]. In Scandinavian conditions, the coefficient of variation, ICC and internal consistency of the ODI is 12%, 0.88-0.91 and 0.94 respectively [71-73]. Good concurrent validity has also been shown [72].
- The EQ-5D measures generic health-related quality of life and is computed into a 0 to 1.00 scale from worst to best possible health state by using the Swedish value sets [74]. A reduction of 0.08 points is considered the MCID in LBP after treatment [75]. Mean change after treatment for LBP has been reported to be 0.12 (SD±0.30) [76].
- The BIPQ analyses cognitive illness representations (consequences, outcome expectancy, personal control, treatment control, and knowledge), emotional representations (concern and emotions) as well as illness comprehensibility. An overall score 0-80 represents the degree to which the LBP is perceived as threatening or benign where a higher score reflects a more threatening view of the illness [52]. The BIPQ has been shown to be valid and reliable in a Scandinavian sample of patients with subacute and chronic LBP. The BIPQ has a Cronbach's alpha =0.72 and a test-retest ICC = 0.86, an ICC range for individual items from 0.64 to 0.88, a standard error of measurement (SEM) = 0.63 and minimal detectable change (MDC) = 1.75[77].
- The PEI has a score range between 0 and 12 with a higher score intended to reflect higher patient self-care enablement [58].
- PGIC asks the patient to rate the degree of change in LBP related problems from the beginning of treatment to the present. This is measured with a balanced 11 point numerical scale. A reduction of 2 points is considered the MCID in LBP after treatment [59].
- PS is measured with a single item patient reported question. The question asks "Over the course of treatment for this episode of low back pain or leg pain, how satisfied were you with the care provided by your health-care provider?" Were you very satisfied (1), somewhat satisfied (2), neither satisfied nor dissatisfied (3), somewhat dissatisfied (4), or very dissatisfied (5)?" [60].

#### Health care process measures:

- At 12 months after baseline, data will also be extracted from the public health care regional registry for the total number of patient visits for LBP, the number patients needing primary care multimodal pain team treatment, the number referred to specialist pain clinic, orthopedic or neurosurgical care and the number receiving surgery.
- Clinical reasoning and process evaluation tool (CRPE-tool): Grade of patient functional impairment and activity limitation according to the ICF brief core set for LBP is assesses by the physiotherapist at baseline and final clinical contact where light, moderate, severe and very severe impairment/limitation is coded 0-4 respectively. A total score for baseline and follow-up measures is calculated from the sum of the functional impairment divided by the number of functional impairments and a similar total score is calculated for activity limitations [61]. ICD-10 diagnosis codes and KVÅ codes for treatment interventions will also be recorded.
- The Keele STarT Back Screening Tool is reported by patients at baseline providing a stratification of prognostic risk of persistent pain. The overall score ranging from 0-9 is used to separate the low risk patients from the medium-risk subgroups where patients who achieve a score of 0-3 are classified into the low-risk subgroup and those with scores of 4-9 into the medium-risk subgroup. To identify the high-risk subgroup, the last 5 items must scoring 4 or 5. The CRPE-tool data will be analysed in terms of StarTback tool subgroups.
- Qualitative SWOT analyses will be performed by HCP between 3-6 months after implementation.
- Semi-structured interviews investigating the patient experience of recieving care for LBP will be performed on 10 patients. These patients will have received care after implementation of the BetterBack<sup>®</sup> model of care.

#### Data management

All paper based questionnaire data will remain confidential and will be kept in a lockable filing cabinet in the research group office. A password-protected coded database only accessible to the research team will be kept on a data storage drive in the research department. The research team will regularly monitor the integrity of trial data. Trial conduct will be audited on a weekly basis by the research team.

#### Statistical analysis

Statistical significance will be assessed with an alpha level of 0.05. All results will be reported as estimates of mean ± standard deviation and also effect size (e.g. mean difference) with 95% confidence intervals (95% CI). An intention-to-treat (ITT) principle applying multiple imputation will be applied. A sensitivity analysis will compare per protocol and ITT databases. A sensitivity analysis will also be used to assess the significance of a washout period by comparing the complete database against the same database without data collected during the 2 weeks in conjunction with the Betterback© implementation in each cluster Matched pairs t-test statistics comparing baseline and follow-up means will be used for the HCP reported primary and secondary outcomes. Causal mediation analysis will be used to analyse indirect mediational effects of multiple putative determinants of implementation behaviour measured with the DIBQ directly after the HCP education and training workshop (intention stage) or at 3 or 12 months (volition stages) on the effect of baseline PCS or PABS-PT on 3 or 12 months follow-up measurement of PCS or PABS-PT. If the HCP education and training workshop does not have a casual effect on improved prospective outcomes we will analyse where the causal pathway breaks down. Causal mediation analysis will be performed using the program PROCESS [81] within IBM SPSS (figure 5).

Patient reported outcome measures for the control and intervention groups will be compared using multilevel analyses of repeated measurements and experiment condition as fixed effects and participants and clusters as random effects with IBM SPSS. Fixed effect interactions between experimental condition and The Keele STarT Back Screening Tool will also be assessed. Patient

population specific minimal clinically important difference will be assessed för primary and secondary outcomes based on an anchor method where PGIC serves as an anchor.

Applying a 1-1-1 multilevel mediation procedure with all effects random in MPLUS, the products of (1) the independent variable (Experimental condition: control or intervention) to the mediator (change in BIPQ), and (2) the mediator to the dependent variable (change in NRS, ODI or secondary outcome scores pre- to posttreatment) when the independent variable is taken into account, will be tested for mediation (figure 6).

The EQ5D will be used to calculate the ratio of costs to quality adjusted life years (QALY) saved for patients. Incremental cost-effectiveness and cost-utility ratios for the multifaceted implementation strategy and the usual care condition will be calculated. This is based on the Swedish guideline priced direct costs of health service utilisation, costs of medications and overall intervention clinical outcome effectiveness and social security system utilisation (sickness benefits) as well as indirect productivity costs due to absenteeism and return to work.

#### **Data monitoring**

All outcome questionnaires are formatted for use of scan processing software for automated data entry into the Statistical Package for the Social Sciences package. The author KS who is not blinded to treatment allocation will perform regular data checks during data entry and provide feedback when necessary to HPC regarding data omissions. JS will also double check data entry to detect and correct input errors, and range checks will be undertaken prior to data analysis.

#### **Ethics and dissemination**

Ethical clearance for the study (Dnr:2017-35/31) has been attained through the Regional Ethics Committee in Linköping.

#### **Internal pilot trial results**

The initial implementation of the BetterBack© model of care in cluster 1 allowed for an internal pilot to determine the HCP acceptability of the intervention and trial within the first cluster [34,35]. A progression criteria for continuing to the main trial required that HCP who have completed the BetterBack© education workshop rate on average a maximum of 2.5 out of 5 on the following determinant of implementation behaviour question: The 27 HCP participating in the internal pilot in cluster 1 responded to the question I expect that the application of BetterBack© model of care will be useful (1 = agree completely - 5 = do not agree at all). A mean value of 1.7 (SD 0.8) was recorded which subsequently fulfilled the HCP progression criteria.

The resulting internal pilot patient flow for april and may were n=28, n=28 for cluster 1 west, n=5, n=12 for cluster 2 central as well as n=14, n=22 for cluster 3 east consecutively. This informed the decision to move cluster 2 central transition from control to intervention condition to occur later in the schedule, planned for september 2017. The flow of patient recruitment and the process of 3 month follow-up in the internal pilot was used to inform the optimal time point of patient reported primary outcome for the main trial. Our initial planning was to measure patient reported primary outcome at 6 months post baseline based on the definition of persistence/chronicity of symptoms being often defined in the literature to be of 3 and up to 6 months duration [82]. However our intern pilot study with a 3 month follow rate of 80% after up to 3 reminders sent to patients informed of a likely risk of non-response at later follow-up time points as patients. Feedback from participating HCP even reported a larger clinical interest in 3 month patient follow-up data. Therefore the internal pilot informed the choice to revise our patient reported primary outcomes to 3 month post-baseline with subsequent amendments of the trial registration on ClinicalTrials.gov: NCT03147300.

Our internal pilot study was also used to assess baseline variation and change over 3 months in HCP

evaluation and patient reported primary outcome measures in the control and intervention arms to aid calibration of the sample size calculation. A multilevel analyses of repeated measurements and experiment condition as fixed effects and participants and clusters as random effects revealed a intracluster correlation of <0.01 for the all primary outcomes measures. Small effect sizes in favour of the intervention condition was shown for PCS (d=0.33) and NRS (d=0.28) primary outcome measures. Therefore, the internal pilot data supported our a priori sample size calculation for the main trial regarding PCS and NRS. However no effect size difference were observed between experimental conditions for ODI. It is possible that when statistical power improves within the main trail, potential differences in ODI may be detectable between experimental conditions.

#### References

- 1. Hoy D, Bain C, Williams G, et al. Systematic review of the global prevalence of low back pain. *Arthritis Rheum* 2012;64:2028-37.
- 2. Hoy D, March L, Brooks P, et al. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. *Ann Rheum Dis* 2014;73:968-74.
- 3. Dionne CE, Dunn KM, Croft PR, et al. A consensus approach toward the standardization of back pain definitions for use in prevalence studies. *Spine* 2008;33:95-103.
- 4. Smart KM, O'Connell NE, Doody C. Towards a mechanisms based classification of pain in musculoskeletal physiotherapy? *Phys Ther Rev* 2008;13:1-10.
- 5. Williams CM, Henschke N, Maher CG, et al. Red flags to screen for vertebral fracture in patients presenting with low-back pain. *Cochrane Database Syst Rev* 2013;1:CD008643.
- 6. Henschke N, Maher CG, Ostelo RW, et al. Red flags to screen for malignancy in patients with low back pain. *Cochrane Database Syst Rev* 2013;2:CD008686.
- 7. Konstantinou K, Dunn KM. Sciatica: review of epidemiological studies and prevalence estimates. *Spine* 2008;33:2464-72.
- 8. Yabuki S, Fukumori N, Takegami M, et al. Prevalence of lumbar spinal stenosis, using the diagnostic support tool, and correlated factors in Japan: a population-based study. *J Orthop Sci* 2013;18:893-900.
- 9. Brinjikji W, Luetmer PH, Comstock B, et al. Systematic literature review of imaging features of spinal degeneration in asymptomatic populations. *Am J Neuroradiol* 2015;36:811-16.
- 10. Wahlin C, Ekberg K, Persson J, et al. Association between clinical and work-related interventions and return-to-work for patients with musculoskeletal or mental disorders. *J Rehabil Med* 2012;44:355-62.
- 11. Nilsing E, Soderberg E, Öberg B. Sickness certificates in Sweden: did the new guidelines improve their quality? *BMC Public Health* 2012;12:907.
- 12. Bernhardsson S, Öberg B, Johansson K, et al. Clinical practice in line with evidence? A survey among primary care physiotherapists in western Sweden. *J Eval Clin Pract*. 2015;21:1169-77.
- 13. National clinical guidelines for non-surgical treatment of newly occurring lumbar nerve root affliction (lumbar radiculopathy), Danish Health Authority; 2016 (In Danish). https://sundhedsstyrelsen.dk/da/udgivelser/2016/lumbal-nerverodspaavirkning-ikke-kirurgisk-behandling. Accessed 03-05-2016.
- 14. National clinical guidelines for non-surgical treatment of newly occurring lower back pain. Danish Health Authority; 2016 (In Danish). https://sundhedsstyrelsen.dk/da/udgivelser/2016/nkr-laenderygsmerter. Accessed 03-05-2016.
- 15. National Clinical Guideline Centre (NICE) Low back pain and sciatica: management of non-specific low back pain and sciatica. Assessment and non-invasive treatments, England; 2016. https://www.nice.org.uk/guidance/indevelopment/gid-cgwave0681/documents. Accessed 03-05-2016
- 16. Thorstensson C, Garellick G, Rystedt H, et al. Better Management of Patients with Osteoarthritis: Development and Nationwide Implementation of an Evidence-Based Supported Osteoarthritis Self-Management Programme. *Musculoskeletal Care*. 2015;13:67-75.

- 17. Skou ST, Roos EM. Good Life with osteoArthritis in Denmark (GLA:D<sup>TM</sup>): evidence-based education and supervised neuromuscular exercise delivered by certified physiotherapists nationwide. BMC Musculoskelet Disord. 2017:18:72.
- 18. Thorstensson C, Dahlberg L, Garellick G. The BOA-register annual report 2014. https://boa.registercentrum.se. Accessed 03-05-2016.
- 19. Skou ST, Roos EM. GLA:D annual report 2015. www.glaid.dk. Accessed 03-05-2016.
- 20. Briggs AM, Jordan JE, Jennings M, et al. A framework to evaluate musculoskeletal models of care. Cornwall: Global Alliance for Musculoskeletal Health of the Bone and Joint Decade; 2016.
- 21. Ajzen I. The theory of planned behavior. Organ Behav Hum Decis Process. 1991;50:179–211.
- 22. Leventhal H, Phillips LA, Burns E. The Common-Sense Model of Self-Regulation (CSM): a dynamic framework for understanding illness self-management. *J Behav Med.* 2016;39:935-46.
- 23. Fixsen DL, Naoom SF, Blase KA, et al. Implementation Research: A Synthesis of the Literature. Tampa, FL: University of South Florida, Louis de la Parte Florida Mental Health Institute. 2005.
- 24. Nilsen P. Making sense of implementation theories, models and frameworks. *Implement Sci* 2015;10:53.
- 25. Nilsen P. (red) Implementering av evidensbaserad praktik. Malmö: Gleerups, 2014.
- 26. Nutley SM, Walter I, Davies HTO. Using Evidence. How Research Can Inform Public Services. Bristol: Policy Press. 2007.
- 27. Eccles MP, Mittman BS. Welcome to Implementation Science. Implement Sci. 2006;1:1.
- 28. Riis A, Elgaard Jensen C, Bro F, et al. A multifaceted implementation strategy versus passive implementation of low back pain guidelines in general practice: a cluster randomised controlled trial. *Implement Sci* 2016;11:143.
- 29. Engers AJ, Wensing M, van Tulder MW, et al. Implementation of the Dutch low back pain guideline for general practitioners: a cluster randomized controlled trial. *Spine* 2005;30:559–600.
- 30. Chan A-W, Tetzlaff JM, Gøtzsche PC, et al. SPIRIT 2013 Explanation and Elaboration: Guidance for protocols of clinical trials. *BMJ* 2013;346:e7586.
- 31. Curran GM, Bauer M, Mittman B, et al. Effectiveness-implementation hybrid designs: combining elements of clinical effectiveness and implementation research to enhance public health impact. *Med Care*. 2012;50:217–26.
- 32. Hooper R, Bourke L. Cluster randomised trials with repeated cross sections: alternatives to parallel group designs. *BMJ* 2015;350:h2925.
- 33. Girling AJ, Hemming K. Statistical efficiency and optimal design for stepped cluster studies under linear mixed effects models. *Statist Med* 2016, 35:2149–66.
- 34. Eldridge S, Kerry S. A practical guide to cluster randomised trials in health service research. Wiley & Sons, 2nd ed, 2012.
- 35. Avery KNL, Williamson PR, Gamble C, et al. Informing efficient randomised controlled trials: exploration of challenges in developing progression criteria for internal pilot studies. *BMJ Open* 2017:7:e013537.
- 36. SBU. Acute neck and back pain: preventive interventions Effects of physical training, manual treatment and cognitive behavioral interventions. Stockholm: Swedish Agency for Health Technology Assessment and Assessment of Social Services (SBU); 2016. SBU report no 245 (in Swedish). http://www.sbu.se/en/publications/sbu-assesses/acute-neck-and-back-pain-preventive-interventions--effects-of-physical-training-manual-treatment-and-cognitive-behavioral-interventions/
- 37. The Swedish National Board of Health and Welfare. National guidelines Methods description. https://www.socialstyrelsen.se/SiteCollectionDocuments/metodbeskrivning-nationella-riktlinjer.pdf . Accessed 03-05-2016.
- 38. GRADE Working Group. Grading quality of evidence and strength of recommendations. *BMJ* 2004;328:1490.

- 39. Slade SC, Kent P, Patel S, et al. Barriers to Primary Care Clinician Adherence to Clinical Guidelines for the Management of Low Back Pain: A Systematic Review and Metasynthesis of Oualitative Studies. *BMC Med Res Methodol* 2017;17:38.
- 40. Jack K, McLean SM, Klaber Moffett J, et al. Barriers to treatment adherence in physiotherapy outpatient clinics: A systematic review. *Man Ther.* 2010;15:220–228.
- 41. Michie S, van Stralen MM, West R. The behaviour change wheel: A new method for characterizing and designing behaviour change interventions. *Implement Sci* 2011;6:42.
- 42. Michie S, Wood CE, Johnston M, et al. Behaviour change techniques: the development and evaluation of a taxonomic method for reporting and describing behaviour change interventions (a suite of five studies involving consensus methods, randomised controlled trials and analysis of qualitative data). *Health Technol Assess* 2015;19:99.
- 43. Cane JE, O'Connor D, Michie S. Validation of the theoretical domains framework for use in behaviour change and implementation research. *Implement Sci* 2012;7:37.
- 44. Michie S, Johnston M, Francis J, et al. From theory to intervention: mapping theoretically derived behavioural determinants to behaviour change techniques. *Appl Psychol* 2008;57:660–680
- 45. Smucker DR, Konrad TR, Curtis P, et al. Practitioner self-confidence and patient outcomes in acute low back pain. *Arch Fam Med* 1998;7:223–8.
- 46. Ostelo RW, Stomp-van den Berg SG, Vlaeyen JW, et al. Health care provider's attitudes and beliefs towards chronic low back pain: the development of a questionnaire. *Man Ther*: 2003, 8:214–22.
- 47. Jensen MP, Turner JA, Romano JM, et al. Comparative reliability and validity of chronic pain intensity measures. *Pain* 1999,83:157-62.
- 48. Chiarotto A, Deyo RA, Terwee CB, et al. Core outcome domains for clinical trials in non-specific low back pain. *Eur Spine J* 201;24:1127–42.
- 49. Clement RC, Welander A, Stowell C, et al. A proposed set of metrics for standardized outcome reporting in the management of low back pain. *Acta Orthop* 2015;86:523–33.
- 50. Fairbank JC, Pynsent PB. The Oswestry disability index. Spine. 2000;25:2940–53.
- 51. EuroQol Group. EuroQol—a new facility for the measurement of health related quality of life. *Health Policy* 1990;16:199–208.
- 52. Broadbent E, Petrie KJ, Main J, et al. The Brief Illness Perception Questionnaire. *J Psychosom Res* 2006, 60:631–37.
- 53. Foster NE, Bishop A, Thomas E, et al. Illness perceptions of low back pain patients in primary care: what are they, do they change and are they associated with outcome? *Pain.* 2008,60:177–87
- 54. Foster NE, Thomas E, Bishop A, et al. Distinctiveness of psychological obstacles to recovery in low back pain patients in primary care. *Pain.* 2010;148:398–406.
- 55. Glattacker M, Heyduck K, Meffert C. Illness beliefs and treatment beliefs as predictors of short-term and medium-term outcome in chronic back pain. *J Rehabil Med.* 2013;45:268–276.
- 56. Campbell P, Foster NE, Thomas E, et al. Prognostic indicators of low back pain in primary care: five-year prospective study. *J Pain*. 2013;14:873–83.
- 57. Løchting I, Garratt AM, Storheim K, et al. The impact of psychological factors on condition-specific, generic and individualized patient reported outcomes in low back pain. *Health Qual Life Outcomes*. 2017,15:40.
- 58. Rööst M, Zielinski A, Petersson C, et al. Reliability and applicability of the Patient Enablement Instrument (PEI) in a Swedish general practice setting. *BMC Family Practice* 2015;16:31.
- 59. Kamper SJ, PT, Maher CG, Mackay G. Global Rating of Change Scales: A Review of Strengths and Weaknesses and Considerations for Design. *J Man Manip Ther* 2009;17:163–70.
- 60. Butler RJ, Johnson WG. Satisfaction with low back pain care. Spine J 2008;8:510–21.
- 61. Cieza A, Stucki G, Weigl M, et al. ICF core sets for low back pain. *J Rehabil Med* 2004;44:69–74.

- 62. Slater H, Davies SJ, Parsons R, et al. A Policy-into-Practice Intervention to Increase the Uptake of Evidence-Based Management of Low Back Pain in Primary Care: A Prospective Cohort Study. *PLoS One*. 2012;7:e38037.
- 63. Tzortziou Brown V, Underwood M, Mohamed N, et al. Professional interventions for general practitioners on the management of musculoskeletal conditions. *Cochrane Database Syst Rev* 2016;6:CD007495.
- 64. Campbell MK, Piaggio G, Elbourne DR, et al. Consort 2010 statement: extension to cluster randomised trials. *BMJ* 2012;345:e5661.
- 65. Mutsaers JHAM, Peters R, Pool-Goudzwaard AL, et al. Psychometric properties of the Pain Attitudes and Beliefs Scale for Physiotherapists: A systematic review. *Man Ther* 2012;17:213-18
- 66. Overmeer T, Boersma K, Main CJ, et al. Do physical therapists change their beliefs, attitudes, knowledge, skills and behaviour after a biopsychosocially orientated university course? J Eval Clin Pract 2009;15:724-732.
- 67. Huijg JM, Gebhardt WA, Crone MR, et al. Discriminant content validity of a Theoretical Domains Framework questionnaire for use in implementation research. *Implement Sci* 2014;9:11.
- 68. Huijg JM, Gebhardt WA, Dusseldorp E, et al. Measuring determinants of implementation behavior: psychometric properties of a questionnaire based on the theoretical domains framework. *Implement Sci* 2014;9:33.
- 69. Childs JD, Piva SR, Fritz JM. Responsiveness of the numeric pain rating scale in patients with low back pain. *Spine* 2005;30:1331–4.
- 70. Ostelo RW, Deyo RA, Stratford P, et al. Interpreting change scores for pain and functional status in low back pain: towards international consensus regarding minimal important change. *Spine* 2008;33:90-4.
- 71. Grotle M, Brox JI, Vøllestad NK. Cross-cultural adaptation of the Norwegian versions of the Roland-Morris Disability Questionnaire and the Oswestry Disability Index. *J Rehabil Med* 2003;35:241-7.
- 72. Lauridsen HH, Hartvigsen J, Manniche C, et al. Danish version of the Oswestry Disability Index for patients with low back pain. Part 1: Cross-cultural adaptation, reliability and validity in two different populations. *Eur Spine J* 2006;15:1705-16.
- 73. Lauridsen HH, Hartvigsen J, Manniche C, et al. Danish version of the Oswestry disability index for patients with low back pain. Part 2: Sensitivity, specificity and clinically significant improvement in two low back pain populations. *Eur Spine J* 2006;15:1717-28.
- 74. Burström K, Sun S, Gerdtham UG, et al. Swedish experience-based value sets for EQ-5D health states. *Qual Life Res* 2014;23:431-42.
- 75. Walters SJ, Brazier JE. Comparison of the minimally important difference for two health state utility measures: EQ-5D and SF-6D. *Qual Life Res* 2005;14:1523–32.
- 76. Soer R, Reneman MF, Speijer BL, et al. Clinimetric properties of the EuroQol-5D in patients with chronic low back pain. *Spine J* 2012;12:1035-39.
- 77. Loechting I, Garratt AM, Storheim K, et al. Evaluation of the brief illness perception questionnaire in sub-acute and chronic low back pain patients: data quality, reliability and validity. *J Pain Relief* 2013;2:122.
- 78. Hill JC, Dunn KM, Lewis M, et al. A primary care back pain screening tool: identifying patient subgroups for initial treatment. *Arthritis Rheum* 2008;59: 632–41.
- 79. Hill JC, Vohora K, Dunn KM, et al. Comparing the STarT Back Screening Tool's subgroup allocation of individual patients with that of independent clinical experts. *Clin J Pain* 2010;26: 783–87.
- 80. Hill JC, Dunn KM, Main CJ, et al. Subgrouping low back pain: a comparison of the STarT Back Tool with the Orebro Musculoskeletal Pain Screening Questionnaire. *Eur J Pain* 2010;14:83–9.

- 81. Hayes AF. PROCESS: A versatile computational tool for observed variable mediation, moderation, and conditional process modeling [White paper]. 2012. Retrieved from http://www.afhayes.com/public/process2012.pdf
- 82. Merskey H, Bogduk N. Classification of chronic pain. 2nd ed. Seattle: IASP Press, 1994. p. 1.

**Authors' contributions:** AA & BÖ formulated the trials original aims and hypothesis. AA, KS, BÖ developed interventions material. AA, KS, PE, PN, ÖB designed the study methodology. AA, KS, PE, PN, ÖB have reviewed and finalised the protocol

**Funding statement:** This work was supported by the Research Council in Southeast Sweden, grant number [FORSS-660371]

**Competing interests statement:** None

Table 1. World health organisation trial registration data set.

| Data category | Information |
|---|---|
| Primary registry and trial identifying | ClinicalTrials.gov |
| number | NCT03147300 |
| Date of registration in primary registry | 03 May, 2017 |
| Prospective Registration: | Yes |
| Secondary identifying numbers | N/A |
| Source(s) of monetary or material support | Linköping University |
| Primary sponsor | Linköping University |
| Secondary sponsor(s) | Simplify and the state of the s |
| Contact for public queries | Allan Abbott, MPhysio, PhD [+46 (0)13 282495] [allan.abbott@liu.se] |
| | Allan Abbott, MPhysio, PhD |
| Contact for scientific queries | Linköping University, Linköping, Sweden |
| Public title | Implementation of a Best Practice Primary Health Care Model for Low Back Pain BetterBack |
| Scientific title | Implementation of a Best Practice Primary Health Care Model for Low Back Pain in Sweden (BetterBack): A Cluster Randomised Trial |
| Countries of recruitment | Sweden |
| Health condition(s) or problem(s) studied | Low back pain |
| \(\frac{1}{2}\) | Behavioral: Current routine practice |
| Intervention(s) | Behavioral: Multifaceted implementation of the BetterBack |
| | Health care practitioner sample |
| | Inclusion Criteria: |
| | - Registered physiotherapists practicing in the allocated clinics and regularly working with patients with LBP |
| | Patient sample |
| | Inclusion Criteria: |
| Key inclusion and exclusion criteria | - Males and females 18-65 years; Fluent in Swedish; Accessing public primary care due to a current episode of a first-time or recurrent debut of benign low back pain with or |
| | without radiculopathy |
| | Exclusion Criteria: |
| | - Current diagnosis of malignancy, spinal fracture, infection, cauda equine syndrome, ankylosing spondylitis or systemic rheumatic disease, previous malignancy during the past 5 |
| | years; Current pregnancy or previous pregnancy up to 3 months before consideration of inclusion; Patients that fulfill criteria for multimodal/multi-professional rehabilitation for |
| | complex longstanding pain; Severe psychiatric diagnosis |
| Study type | Interventional |
| Date of first enrolment | April 1, 2017 |
| Target sample size | 600 |
| Recruitment status | Recruiting |
| | - Incidence of participating patients receiving specialist care [Time Frame: 12 months after baseline] |
| Primary outcome(s) | - Numeric rating scale (NRS) for lower back related pain intensity during the latest week [Time Frame: Change between baseline and 3 months post baseline] |
| | - Oswestry disability index (ODI) version 2.1 [Time Frame: Change between baseline and 3 months post baseline] |
| | - Practitioner Confidence Scale (PCS) [Time Frame: Change between baseline and 3 months post baseline] |
| | - Clinician rated health care process measures [Time Frame: Baseline and final clinical contact (Up to 3 months where the time point is variable depending upon the amount of |
| | clinical contact required for each patient)] |
| | - Numeric rating scale (NRS) for lower back related pain intensity during the latest week [Time Frame: Baseline, 3, 6 and 12 months] |
| | - Oswestry disability index (ODI) version 2.1 [Time Frame: Baseline, 3, 6 and 12 months] |
| V ay aaaan dawy ay taamaa | - Pain Attitudes and Beliefs Scale for physical therapists (PABS-PT) [Time Frame: Baseline, directly after education and at 3 and 12 months afterwards] |
| Key secondary outcomes | - Patient Enablement Index (PEI) [Time Frame: 3, 6 and 12 months] - Patient global rating of change (PGIC) [Time Frame: 3, 6 and 12 months] |
| | - Patient global rating of change (PGIC) [Time Frame: 3, 6 and 12 months] - Patient satisfaction [Time Frame: 3, 6 and 12 months] |
| | - Practitioner Confidence Scale (PCS) [Time Frame: Baseline, directly after commencement of implementation strategy and at 3 and 12 months afterwards] |
| | - Practitioner Confidence Scale (PCS) [Time Frame: Baseline, directly after commencement of implementation strategy and at 3 and 12 months afterwards] - The Brief Illness Perception Questionnaire (BIPQ) [Time Frame: Baseline, 3, 6 and 12 months] |
| | - The European Quality of Life Questionnaire (EQ-5D) [Time Frame: Baseline, 3, 6 and 12 months] |
| | - The European Quanty of Life Questionnaire (EQ-3D) [Time Frame: Basenire, 3, 6 and 12 months] |

*Table 2. Study design and schedule of enrolment, interventions and assessments* 

| | Table 2. Study | | | U | | | | | | | | | , | , | | 1 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Tir | neline | June 2016<br>- Feb 2017 | Mar 2017 | Apr 2017 | May 2017 | Jun 2017 | Jul 2017 | Aug 2017 | Sep 2017 | Oct 2017 | Nov 2017 | Dec 2017 | Jan 2018 | Final clinic<br>visit | Follow-up<br>3 months<br>after<br>baseline | | |
| En | rolment schedule | | HCP Cluster | cruitment | | ı | Patient re | | | | | | | | | | |
| | | | random | during into | | | | | | 8 | P | | | | | | |
| | | | allocation | pha | | | | | | | | | | | | | |
| Intervention schedule | | MOC and protocol development | Cluster 1<br>West | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | 1 | | | | |
| | | | internal pilot | | | | | | | | | | | | | | |
| | | | Cluster 2<br>Central | 0 | 0 | 0 | 0 | MOC implementation | 1 | 1 | 1 | 1 | 1 | | | | |
| | | | Cluster 3<br>East | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0<br>MOC<br>implementation | | | | |
| Ass | sessment schedule | | | Baselir | | | | | | ne data | | | | | l measures ir | | |
| | | | | Internal p | ilot (T=0) | | | | Main tr | ial (T=0) | | | T | (T=1) | (T=2) | ( T=3) | (T=4) |
| ntation | PCS | | Cluster 1<br>before and after<br>MOC<br>implementation | | | | | Cluster 2<br>before and after<br>MOC<br>implementation | | | | | Cluster 3<br>before and after<br>MOC<br>implementation | | х | | х |
| HCP implementation | PABS-PT | | Cluster 1<br>before MOC<br>implementation | | | | | Cluster 2<br>before MOC<br>implementation | | | | | Cluster 3<br>before MOC<br>implementation | | Х | | х |
| | DIBQ | | Cluster 1<br>after MOC<br>implementation | | | | | Cluster 2<br>after MOC<br>implementation | | | | | Cluster 3<br>after MOC<br>implementation | | Х | | Х |
| | NRS back pain and leg pain | | | Х | Х | Х | Х | Х | Х | Х | Х | х | Х | | Х | Х | Х |
| | ODI | | | Х | Х | Х | Х | X | Х | Х | Х | Х | Х | | Х | Х | Х |
| <b>PROMS</b> | EQ5D | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | х | | Х | Х | Х |
| 8 | BIPQ | | | Х | Х | Х | Х | Х | Х | Х | Х | Х | Х | | Х | Х | Х |
| ۵ | PEI | | | | | | | | | | | | | | Х | Х | Х |
| | Patient satisfaction | | | | | | | | | | | | | | Х | Х | Х |
| | PGIC | | | | | | | | | | | | | | Х | Х | Х |
| Process | HCP assessment,<br>diagnosis and<br>treatment of<br>patients | | | х | х | х | х | х | х | х | х | х | х | х | | | |
| | Referrals to specialist care | | | | | | | | | | | | | | | | Х |

MOC=model of care, 0=Control condition, 1=Intervention condition, PROMS=Patient reported outcome measures, grey shaded cells=internal pilot, T= assessment time. Period where 2 week cross-over from control to intervention can occur dependent upon patient recruitment rates identified in the internal pilot study.

Table 3. Characterizing the BetterBack© model of care intervention content and mechanisms of action using the behaviour change wheel [41], Behavioural change technique (BCT) taxonomy (v1) [42], and the TDF [43].

| Target | Rationale based on | В | etterBack© Intervention content | Mech | anism of action | | |
|---|---|---|---|---|---|---|---|
| behavior | barriers to be addressed | Mode | Content | BCT[42] | Functions | COM-B | TDF |
| Improved HCP | 1) Low beliefs about | 1) Workshop | Evidence based model of care and | 1.2 Problem-solving | Enablement | Psychological capability | Behavioral regulation |
| confidence and | skills/capabilities for | lls/capabilities for clinical implementation tools (S | | 1.4 Action planning | Enablement | Psychological capability | Goals |
| | improving self-care patient | | supplementary files 1 & 2) | 2.2 Feedback on behaviour | Training | Reflective motivation | Behavioral regulation |
| orientation in | management | | | 3.1 Social support | Enablement | Social opportunity | Social Influences |
| treating LBP through | 2) Use of a biomedical treatment orientation rather | | | 4.1 Instruction on how to perform behaviour | Education | Psychological capability | Knowledge |
| adoption of<br>BetterBack© | than a biopychosocial orientation | | | 5.3 Information about social and environmental consequences | Persuasion | Social opportunity<br>Physical opportunity | Social Influences Environmental context and resources |
| model of care | 3) Low awareness of the | | | 6.1 Demonstration of behaviour | Modelling | Psychological capability | |
| | model | | | 6.2 Social comparison | Persuasion | Social opportunity | Social Influences |
| | 4) Beliefs of negative consequences of the model | | | 6.3 Information about other's approval | Persuasion | ** | Social Influences |
| | | | | 8.1 Behavioural practice/rehearsal | Training | Physical capability | Physical skills |
| | | | | 8.7 Graded task | Training | Physical capability | Physical skills |
| | | | | 9.1 Credible source | Persuasion | | Reinforcement |
| | | | | 9.2 Pros and cons | Persuasion | | Beliefs about Consequences |
| | | | | 9.3 Comparative imagining of future outcomes | Enablement | Reflective motivation | Beliefs about Consequences |
| | | | | 13.2 Framing/reframing | Enablement | Psychological capability | Cognitive and interpersonal skills |
| | | | | 15.1 Verbal persuasion about capability | Enablement | Psychological capability<br>Physical capability | Beliefs about capabilities |
| | | 2) Report and website | Evidence based model of care and clinical implementation tools (See | 4.1 Instruction on how to perform | Education | Psychological capability | Knowledge |
| | | dissemination | supplementary file 2) | 6.3 Information about other's approval | Persuasion | Social opportunity | Social Influences |
| Decreased patient LBP and | 1) Maladaptive beliefs on the cause and course of LBP | | , , , , , , | 5.1 Information about health consequences | Education | Psychological capability | Knowledge |
| disability as<br>well as<br>improved<br>patient | outcome expectation,<br>anxiety, catastrophizing,<br>fear-avoidance, illness | | | 9.1 Credible source | Persuasion | Reflective motivation | Reinforcement |
| enablement of self-care | beliefs. | 2) BetterBack©<br>Part 1. Patient | Lay language education on the spine's structure and function, | 4.1 Instruction on how to perform behaviour | Education | Psychological capability | Knowledge |
| | | education<br>brochure | natural course of benign LBP and advice on self-care | 5.1 Information about health consequences | Education | Psychological capability | Knowledge |
| | ability to perform activities, | 3) BetterBack© | Pain physiology, biomechanics, | 1.2 Problem-solving | Enablement | Psychological capability | Behavioral regulation |
| | low baseline physical | Part 2. Group | | 3.1 Social support | Enablement | | Social Influences |
| | activity. | education | | 4.1 Instruction on how to perform | Education | Psychological capability | Knowledge |

| | | behaviour | | | |
|---|---|---|---|---|---|
| | | 4.3 Re-attribution | Education | Psychological capability | Knowledge |
| | | 5.1 Information about health | Education | Psychological capability | |
| | | consequences | | , , , | |
| | | 6.1 Demonstration of behaviour | Modelling | Psychological capability | Social Influences |
| | | 6.2 Social comparison | Persuasion | Social opportunity | Social Influences |
| | | 8.1 Behavioural practice/rehearsal | Training | Physical capability | Physical skills |
| | | 8.2 Behaviour substitution | Enablement | Psychological capability | Behavioral regulation |
| | | 9.1 Credible source | Persuasion | Reflective motivation | Reinforcement |
| | | 9.3 Comparative imagining of future outcomes | Enablement | Reflective motivation | Beliefs about Consequences |
| | | 10.8 Incentive (CME diploma) | Enablement | | Reinforcement |
| | | 11.2 Reduce negative emotions | | Reflective motivation | Emotion |
| | | 12.4 Distraction | Enablement | | Memory, attention and decision |
| | | | | | processes |
| | | 12.6 Body changes | Training | | Physical skills |
| | | 13.2 Framing/reframing | | | Cognitive and interpersonal skills |
| 4) BetterBack@ | | 1.1 Goal-setting | Enablement | | Goals |
| Part 1. | modulation strategies and | 1.5 Review behaviour goal(s) | Enablement | | Goals |
| Individualised | functional restoration strategies. | 2.2 Feedback on behaviour | | | Behavioral regulation |
| physiotherapy | Treatment matched to patient | 6.1 Demonstration of behaviour | | Psychological capability | |
| | specific functional impairment and activity limitations. | 7.1 Prompts/cues | Environmental | | Environmental Context and Resources |
| | Individualised dosing. | 8.1 Behavioural practice/rehearsal | restructuring | II. | Physical skills |
| | marviadansea desing. | 8.7 Graded task | | | Physical skills |
| | | 9.1 Credible source | Persuasion | J 1 J | Reinforcement |
| | | | | | Physical skills |
| | | 12.6 Body changes | Training | | |
| | | 15.1 Verbal persuasion about capability | | Physical capability | Beliefs about capabilities |
| | Patient mediated self-care pain | 1.1 Goal-setting | Enablement | | Goals |
| | | 1.5 Review behaviour goal(s) | Enablement | | Goals |
| home based | restoration strategies and general | 1.8 Behavioural contract | Incentivisation | | Intentions |
| physiotherapy | exercise. Treatment matched to patient specific functional | 2.3 Self-monitoring of<br>Behaviour (Training diary) | Training | | Behavioral regulation |
| | impairment and activity | 2.2 Feedback on behaviour | Training | | Behavioral regulation |
| | limitations. Individualised dosing. | 3.1 Social support | Enablement | Social opportunity | Social Influences |
| | | 6.1 Demonstration of behaviour | Modelling | Psychological capability | Social Influences |
| | | 6.2 Social comparison | Persuasion | | Social Influences |
| | | 8.1 Behavioural practice/rehearsal | Training | | Physical skills |
| | | 8.7 Graded task | Training | Physical capability | Physical skills |
| | | 9.1 Credible source | Persuasion | Reflective motivation | Reinforcement |
| | | 12.6 Body changes | Training | | Physical skills |
| | | 15.1 Verbal persuasion about | Enablement | Psychological capability | Beliefs about capabilities |

Figure 1. Municipal resident population and number of physiotherapy rehabilitation clinics and therapists in the west, central and east organisational clusters in Östergötland health care region



Figure 2. Current routine care clinical pathway for LBP in Östergötland health care region. The primary care physiotherapy process outlined by the red square is the focus area for the implementation of the BetterBack@model of care for LBP



Figure 3. The Behavioral Change Wheel



Policy categories



Intervention functions



#### **TDF** domains

Soc - Social influences

Env - Environmental Context and Resources

Id - Social/Professional Role and Identity

Bel Cap - Beliefs about Capabilities

Opt - Optimism

Int - Intentions

Goals - Goals

Bel Cons - Beliefs about Consequences

Reinf - Reinforcement

Em - Emotion

Know - Knowledge

Cog - Cognitive and interpersonal skills

Mem - Memory, Attention and Decision Processes

Beh Reg - Behavioural Regulation

Phys - Physical skills



Sources of behaviour



Figure 4. BetterBack@model of care for LBP



Figure 5. Causal mediation model to analyse indirect mediational effects  $(a^k b^k)$  of multiple putative determinants of implementation behaviour measured with the DIBQ directly after the HCP education/training workshop (intention stage) or at 3 or 12 months (volition stages) for the effect of baseline PCS or PABS-PT on 3 or 12 months follow-up measurement of PCS or PABS-PT (c').



Figure 6. 1-1-1 multilevel mediation model with all variables measured at level-1 but all causal paths (direct= $c_j$ ', indirect= $a_jb_j$ , and total effects= $c_j$ '+  $a_jb_j$ ) are allowed to vary between level-2 clusters.



#### Supplementary file 1

## Östergötland health care region physiotherapeutic clinical practice guideline recommendations for primary care management of benign LBP with or without radiculopathy

Each evidence based guideline recommendation is supported by a clinical priority ranking. This is based on an overall assessment of the severity of the condition, reported effect of the intervention, strength of evidence assessment (GRADE), cost-effectiveness and the benefit of the intervention based on professional experience and patient benefit. A scale from 1 to 10 is used where the number 1 indicates recommended practices with the highest priority while the number 9 indicates recommended practices of low priority. The number 10 indicates recommendations that provide very little or no benefit or utility and are therefore not recommended.



**Recommendation 1** 

PRIORITY RANKING = 12345678910

Routine care should consist of standardised processes for subjective and objective assessment and diagnostics. A thorough screening of red flags is essential to rule out serious pathology. Treatment should be individualised for each patient. Basic treatment principles should be based on reassurance of a good prognosis, maintenance of appropriate physical activity and self-care enablement.

Justification: The work group's reasoning is based on clinical experience of the importance of careful screening to rule out serious pathology. Furthermore, standardised assessment and diagnostics provide quality assurance but treatment needs to be individualised for each patient case. The work group also reasoned based on clinical experience that appropriate physical activity is likely to contribute to maintaining the patient's functional level, psychosocial and general health as well as have positive effects on self-care enablement. In some cases, may physical activity temporarily aggravate pain and symptoms, but there are no known persisting side effects. The work groups reasoning is also based on evidence showing a statistically significant advantage for maintaining appropriate physical activity compared to bed rest for improving pain and function. Despite this, evidence that proves the benefit of appropriate physical activity is so great to be clinically relevant is missing. In addition, the best available evidence has however a currently limited scientific basis ( $\otimes\otimes\circ\circ$ ). The working group proposes the following resources in the BetterBack model of care to support the implementation of Recommendation 1 (See sections 7.1-7.5)

**Recommendation 2** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

Do not perform routine medical imaging investigations (eg X-ray, CT, MRI)

Justification: The work group's reasoning is based on evidence that shows no differences in outcomes of pain, function and quality of life between patients who received or did not receive routine medical imaging investigations in the primary care context. The best available evidence has however a currently inadequate scientific basis ( $\otimes$ OOO). It was also discussed that imaging cannot confirm or reject a preliminary diagnosis as the relationship between patient symptoms and degenerative imaging finding is usually weak. Moreover, degenerative secondary findings are common in asymptomatic individuals. *The work group however suggests that early use of medical imaging is motivated in the presence of symptoms or signs suggesting possible serious underlying pathology (red flags). Medical imaging may also be relevant when pain persists despite primary care treatment.* 

**Recommendation 3** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

Consider using a patient-reported tool (eg STarT Back risk assessment tool) as usual care during the early-stages of patient management to screen the risk of continued LBP Justification: The work group's reasoning is based on studies showing that STarT Back Tool is the only valid tool to investigate the risk of continued back pain in the primary care context. It shows the highest accuracy for detecting patients with low risk profile (total score  $\leq$ 3) and medium-high risk profile (total score  $\geq$ 4) for continued back pain. Studies also show that STarT Back Tool has the best ability to predict functional and pain-related outcomes. The best available evidence has however a currently inadequate scientific basis ( $\otimes$ 000). No economical evaluations were identified but the working group discussed the importance of a simple and fast tool. STarT Back Tool can be filled in and analyzed in a few minutes to advantage over other tools that can be an administrative burden for patients and healthcare professionals. The working group argues that the predictive value of the tool should support, but not replace, regular examination procedures and clinical decision making. See section 7.3 for STarT Back Tool.

**Recommendation 4** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

Consider using a patient-reported tool (such as the STarT Back risk assessment tool) and classification of examination findings during the early-stages of patient management to aid the stratification of care to prevent continued LBP

Justification: The work group reasoned that for the choice and scope of targeted treatment measures, consideration should be given to the assessment of risk profile for long-term LBP and classification of examination findings. This has been shown to have a better effect on pain, function and quality of life, as well as less economic costs compared to no treatment stratification. The best available evidence has however a currently inadequate scientific basis ( $\otimes$ OOO). For a patient with low risk profile (total score  $\leq$ 3 on STarT Back Tool) usual care is relevant and requires only few visits, but the working group recommends that adequate treatment measures directed at examination findings is of the highest importance. For patients with medium-high risk profile (total score  $\geq$  4 on STarT Back Tool), usual care will require additional visits. Information provided in questions 5-9 on STarT Back Tool that investigate anxiety with psychological risk factors can guide the need, focus and extent of behavioral medicine measures. The working group arques that stratified care classified after assessing a risk profile for long-term back pain should

support but not replace conventional examination procedures and clinical decision-making for treatment measures. The working group proposes the following resources to support the implementation of targeted treatments based on stratification (See sections 7.1-7.5).

**Recommendation 5** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10













Consider giving individualised patient education as a part of usual care (e.g. an explanatory model based on pain neuroscience and psychological mechanisms)

Justification: Based on the best available evidence, the work group reasoned that individualised patient education as part of usual care can result in reduced work sickness absenteeism. The priority of the recommendation has been strengthened by consensus within the work group based on proven experience that individual adapted patient education is an important part of patient-centered care. The best available evidence has however a currently inadequate scientific basis ( $\otimes \circ \circ \circ$ ). The intervention requires that the patient is receptive for education. The extent of patient education can depend upon whether the patient has a distorted image of the underlying mechanism of LBP and a high degree of negative outcome expectations, anxiety, and fear-avoidance or if they are inactive or passive in managing the LBP. Patient education should include a reassuring dialogue and other cognitive and behavioural therapeutic techniques of relevance to support change in the individual's maladaptive thoughts, feelings and behaviors. Pedagogical explanation models should be used to provide the patient with knowledge about symptoms and disorders, as well as to strengthen and support self-care ability to master everyday activities. The work group proposes the following resources to support of the implementation of patient education (See sections 7.6-7.7)

**Recommendation 6** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10













#### Consider a supervised exercise program as part of usual care

Justification: Supervised training is defined as general or back-specific exercises or physical activities conducted under the guidance of a healthcare professionals. The work group's reasoning is based on scientific evidence and proven experience that supervised training as part of usual care can result in clinically relevant improvement in pain, function, quality of life and produces lower health care costs compared with no supervised training. There is however no evidence that a specific type of exercise would be superior to another. The best available evidence has however a currently limited scientific basis ( $\otimes \otimes \circ \circ$ ). The work group proposes the following resources to support the implementation of a supervised training program (see section 7.8).

**Recommendation 7** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10













Consider mobilisation techniques for neuromusculoskeletal structures as part of usual care (including active or passive motion in an angular and / or translational plane) Justification: The working group reasoning is based on evidence that for patients with segmental movement impairments, mobilization techniques can provide a statistically significant reduction in short-term pain. It is however uncertain whether the effect is sufficiently large so that patients experience a clear improvement overtime. At group level, there is no evidence that a particular technique is be superior to another. It cannot be

ruled out that for subgroups of LBP patients, more positive effects on pain and function may be produced by specific mobilisation techniques. It is expected that these subgroups can be identified by careful diagnostics and short trial treatments. Mobilizing techniques as part of multimodal treatment provide better results. Serious side effects are rare. However, the best available evidence is based on a currently limited scientific basis  $(\otimes \otimes \circ)$ .

**Recommendation 8** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

#### Consider acupuncture treatment in addition to usual care

Justification: The working group reasoned based on evidence that cannot exclude acupuncture has a short-term pain relief effect in addition to a placebo effect. Acupuncture has however no effect on function. Side effects in the form of brief superficial bleeding or inflammation may occur. Pneumothorax and systemic infections are not common, but the prevalence is unknown. The best available evidence has however a currently inadequate scientific basis ( $\otimes \circ \circ$ ).

**Recommendation 9** 

PRIORITY RANKING = 12345678910

#### Do not offer corset, shoes, traction, ultrasound or electrotherapy

Justification: The work group's reasoning is based on evidence that passive treatments such as corset, shoots / soles, traction, ultrasound or electrotherapy do not reduce pain or improve function and quality of life in patients more than no treatment or when offered as part of multimodal treatment. However, the best available evidence is based on a currently limited scientific basis ( $\otimes\otimes\bigcirc\bigcirc$ ). It cannot be ruled out that subgroups of patients may experience positive effects of these interventions when a hypothesised effect mechanism is aimed at specific functional impairment or activity limitation.

**Recommendation 10** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

### Consider prescription-free NSAID medication if necessary in addition to usual treatment (lowest dose and shortest possible treatment time).

NSAIDs: There is evidence of the effect of NSAID in patients with long-term LBP but the effect has not been highlighted on short-term pain or functional outcomes. There are no adverse reactions reported in systematic review studies on LBP, but potential transient side effects of NSAIDs such as reduced blood clotting, reduced stomach mucous function and reduced kidney function are known from studies on other conditions. The work group reasoned that lowest dose and shortest possible treatment time decreases the risk of side-effects. The work group anticipates that there are differences in patient preferences regarding NSAIDs, where some patients will agree to NSAID treatment, while others will decline. The best available evidence for NSAID effects on LBP outcomes is based on an inadequate scientific evidence ( $\otimes \circ \circ \circ$ ). The work group reasoned based on clinical experience that it cannot be excluded that the NSAID may have a pain relief effect in the short term.

**Recommendation 11** 

PRIORITY RANKING = 1 2 3 4 5 6 7 8 9 10

#### Do not offer paracetamol or opioids

Paracetomol: Has no effect on the degree of LBP and functional ability. There are no reported adverse reactions in studies, but side effects of paracetamol in the form of hepatic effects are known from studies on other conditions. The best available evidence is based on a moderately strong scientific basis ( $\otimes\otimes\otimes\circ$ ).

Opioids: A weak analgesic effect of oxycodone in combination with paracetamol has been demonstrated in a study but the intervention has no effect on functional capacity for up to 12 weeks. Other positive effects or adverse effects were not shown. A wide range of opioid side effects are known from other studies. Therefore, the working group reasoned that treatment results in more risks than benefits to the patient. The best available evidence is based on a currently limited scientific basis ( $\otimes\otimes$ ).

Implementation support tools
1. Subjective assessment proformer for therapist use

| LOW BACK SUBJECTIVE ASS | SESSMENT PROFOI | RMER | |
|---|---|---|---|
| Name: Date of birth: | | | |
| Date: | la | | |
| History of the present condition (debut, duration, activity limitation) | Symptom localisation | | |
| Symptom Description | Localisation back | Localisation right leg | Localisation<br>left leg |
| Pain nature (Dull, stabbing, radiating etc) | | | |
| Pain frequency (Constant/ Intermittent) | | | |
| Pain Intensity (NRS 0-10) | | | |
| Daily variation (am/pm, night time pain/disturbed sleep) | | | |
| Irritability (non-irritable/highly irritable) | | | |
| Aggravating factors (loading etc) | | | |
| Easing faktors (rest etc) | | | |
| Course (Improving/same/worse) | | | |
| Other symptoms (Instability, weakness, paresthesia, stiffness) | | | |
| Past medical history Previous level of function/activity: | Red flags: (malignancy, unexplained weight loss, trauma, osteoporosis, infection, inflammatory disease, spinal cord compression symtoms, drug use) | | |
| Previous treatment: | Other illnesses/ General health: | | |
| Work, Social, Family history | Patient förväntnir | ngar | |
| Medication | Medical imaging/ | Laboratory tests | |

2. Physical assessment proformer

| | | | | | | | | | L | ow | BA | CK P | PHYS | SICA | ۱L A | SSESSMENT P | ROF | FORM | ИER | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| 1. INSPEC | 1. INSPECTION – Postural screen Sitting: good/fair/poor Postural correction: Bette | | | | | | | | | | | | | | | | | | | | | | | | | | | | | | |
| Sitting: g | ood/fa | ir/p | oor | | | | | | | Pc | stur | al c | orre | ctic | n: E | etter/Worse/ | No ( | effec | t | | | | | | | | | | | | |
| Standing | : good/ | fair, | /poc | r | | | | | | Pc | stur | al c | orre | ctic | n: E | Better/Worse/No effect | | | | | | | | | | | | | | | |
| Lordosis | Lordosis: Hyper/hypo/normal Kyphosis: Hyper/hypo/ | | | | | | | | | | | | | | o/normal Lateralt shift: Right/Left/none | | | | | | | | | | | | | | | | |
| Spinal sy | mmetr | y: | | | | | | | | Sh | ould | ler s | sym | me | try: | Pelvic symmetry: | | | | | | | | | | | | | | | |
| Leg & fot | Leg & fot symmetry: Muscular hypo/hyperti | | | | | | | | | | | | | | rtrophy: Scars: | | | | | | | | | | | | | | | | |
| | | | | | | | | | | | | 3. SCREENING TEST IN STANDING/SITTING | | | | | | | | | | | | | | | | | | | |
| | Shoes on/off, sit-stand, 2 leg/ 1 leg squat, lunge right/left | | | | | | | | | | | | | | | | | | | | | Rig | ght | | | Let | ft | | | | |
| Gait: Trer | ndelenk | ourg | righ | ıt/le | ft | | | | | | | | | | | Slump test | + se | nsitis | satio | n | | | | | | | | | | | |
| | p right, | | | | | | | | | | | | | | | head/foot | | | | | | | | | | | | | | | |
| | ight tra<br>walkin | | _ | | eft | | | | | | | | | | | Foramen co | mpi | ressi | on/ເ | unloa | adin | g | | | | | | | | | |
| | el walki | ng r | ight/ | | | | | | | | | | | | | Hip loading | /unl | loadi | ng i | n sta | ndi | ng | | | | | | - | | | |
| | | | | <b>TINI</b> | | | | | | | | | _ | | | F TEST IN S | IDE | 13/151 | _ | | | | | | | | | 丄 | | | |
| 4. TEST IN LUMBAR A | | | | | | /EN/I | NIT | | | | | | | | | 5. TEST IN S<br>LUMBAR PA | | | | II A D | N// | \\/ER | MEN | т | | | | | | | |
| LUIVIDAN | Range | | GUL | AN I | VIOV | Qua | | | | Cvr | npto | mc | | | | LOIVIDAR PA | 1 | | VGC | LAN | IVIC | JVEI | _ | mpt | om | | | | | | |
| | Nalige | 1 | | 1 | | Qua | пц | | | | ring | _ | <u>ا</u> | Re | | - | Nai | nge | 1 | | 1 | | <u> </u> | | _ | nd | | Dor | | Ov | ٥.۲ |
| | Large | M | led | Sm | all | High | 1 | Low | ' | | ririg<br>ige | | u<br>ige | M | • | | Lar | ge | Me | ed | Sm | all | | ıring<br>nge | | nu<br>ange | | Rep<br>Mo | | pre | |
| Flex | | | | | | | | | | | | | | | | Flex | | | | | | | | | | | | Ì | | | |
| Ext | | | | | | | | | | | | | | | | Ext | | | | | | | | | | | | | | | |
| Lateral | | 1_ | | 1_ | | | | | _ | | | <u> </u> | | | | Lat | R | L | R | L | R | L | R | L | F | ٦ L | L | R | L | R | L |
| flex | R L | R | L | R | L | R | L | R | L | R | L | R | L | R | L | flex | _ | | R | | | | _ | | | | | _ | | | |
| Side<br>Glide | R L | R | L | R | L | R | L | R | L | R | L | R | L | R | L | Rot | R | | | | | L | | L | | R L | | R | | R | |
| Rot | R L | R | L | R | L | R | L | R | L | R | L | R | L | R | L | Coupled<br>flex | R | L | R | L | R | L | R | L | F | R L | L | R | L | R | L |
| Coupled<br>flex | R L | R | L | R | L | R | L | R | L | R | L | R | L | R | L | Coupled ext | R | L | R | L | R | L | R | L | F | R L | L | R | L | R | L |
| Coupled ext | R L | R | L | R | L | R | L | R | L | R | L | R | L | R | L | | | | | | | | | | | | | | | | |
| 6. PRONE | | - ! | | | | | | | | | | - | | | | 7. SUPINE | | | | | | | | | | | | | | | |
| ACCESSOR | RY MON | /EM | ENT | /NE | RVE | & IV | IUS | CLE | FU | NCT | ION | | | | | DIFFERENTI | AL C | DIAG | NOS | TICS | н | P/SI- | IOI | NT/E | BAC | K | | | | | |
| Spinal ext | | | | | | | _ | | _ | | se/N | | ffec | t | | Spinal flexion | | | | | | • | | Bett | | | rse | /No | effe | ct | |
| Segmenta | | | | | | | | | _ | | ent | | | Pai | n | Isometric/d | | | | omin | al | | | | | | | | | | |
| | · | | | | | | Н | lypei | · Н | уро | Nor | mal | | | | muscle test | S | | | | | | | | | | | | | | |
| - Central F | P/A, Sp | ring | ing t | est | | | | | | | | | | | | | | | | | | | | ı | Righ | nt | | | Le | ft | |
| - Unilatera | al P/A | | | | | | | | | | | | | | | Hip: Angula | r mo | oven | nent | | | | | | | | | $\top$ | | | |
| - Rotation | provo | catio | on | | | | | | | | | | | | | Patricks tes | | | | , | | | | | | | | | | | |
| - Prone in | stabilit | y tes | st | | | | | | | | | | | | | SI-joint prov | _ | | | , ASI | LR | | | | | | | | | | |
| Femoral n | erve te | nsic | on te | st | | | | | | | | | | | | <b>∭</b> ′ ′ | | | | • | | | | | | | | | | | |
| | | | | | | | | | | | | Passive SLR | + he | ead/ | foot | | | | | | | | | | | | | | | | |
| Isometric | /dynam | nic b | ack | mus | cle | | | | | | | | | | | sensitisatio | n, cr | rosse | d SL | .R | | | | | | | | | | | |
| tests | | | | | | | | | | | | | | | | Myotomes- | L1- | 2(I), | <b>L2</b> -3 | s(Q), | | | | | | | | | | | |
| | | | | | | | | | | | | | | | | ,<br>L4-5(TA), L5 | | | | | 1(TS | 5) | | | | | | | | | |
| 8. PALPAT | ION | | | | | | | | | | | | | | | Dermatome | es | | | | | | | | | _ | | | | | |
| | | | | | | | | | | | | | | | | Reflexs: Pat | ella | L3-4 | , Ac | hilles | s S1 | | | | | | | $\dagger$ | | | |
| | | | | | | | | | | | | | | | | Babinski, Kl | onu | S | | | | | | | | | | $\dagger$ | | | |
| l | | | | | | | | | | | | | | | | II | | | | | | | | | | | | | | | |

#### 3. STarT Back Tool

| | Patient name: | | | Date: | | | |
|---|---|---|---|---|---|---|---|
| | Thinking about the | last 2 weeks tio | k your response to | the following quest | tions: | Disagree | Agree |
| 1 | My back pain has sp | 5 | | | | | |
| 2 | I have had pain in th | | | | | | |
| 3 | 3 I have only walked short distances because of my back pain | | | | | | |
| 4 | 4 In the last 2 weeks, I have dressed more slowly than usual because of back pain | | | | | | |
| 5 | It's not really safe fo | | | | | | |
| 6 | Worrying thoughts | | | | | | |
| 7 | I feel that my back p | pain is terrible | and it's never goin | ig to get any better | r | | |
| 8 | In general I have no | t enjoyed all th | e things I used to en | ijoy | | | |
| 9. | Overall, how bother | some has your l | oack pain been in th | ie last 2 weeks? | | | |
| | Not at all | Slightly | Moderately | Very much | Extre | nely | |
| | 0 | 0 | 0 | □<br>1 | 1 | | |
| | Total score (all 9): | | Sub Scor | re (Q5-9): | | | |

© Keele University 01/08/07 Funded by Arthritis Research UK

4. Clinical Reasoning and Process Evaluation tool (CRPE-tool) for therapists
| PATIENT NAME: | First assessment date:// |
|----------------|----------------------------------------|
| DATE OF BIRTH: | Final assessment date:// |
| DATE OF BIRTH. | Totalt number of physiotherapy visits: |

### **ASSESSMENT**

- First assessment cross X relevant assessment findings
- $\bullet \quad \hbox{Final assessment circle } \bigcirc \ \hbox{relevant assessment findings}$

| | | | | | | KVÅ |
|---|---|---|---|---|---|---|
| 1. Assess grade of <u>FUNCTIONAL IMPAIRMENT</u> | None | Lite | Moderate | Severe | Complete | code |
| Energy and drive (motivation) | 0 | 1 | 2 | 3 | 4 | PA006 |
| Sleep functions | 0 | 1 | 2 | 3 | 4 | PA007 |
| Emotional functions (anxiety, low mood) | 0 | 1 | 2 | 3 | 4 | PA011 |
| Thought functions (physical symptoms caused by | 0 | 1 | 2 | 3 | 4 | PA013 |
| cognitive/rational factors) | | | | | | |
| Sensory function (sensitivity for pain "sensitisation") | 0 | 1 | 2 | 3 | 4 | PB008 |
| Pain (choose relevant category) | | | | | | |
| Back pain | 0 | 1 | 2 | 3 | 4 | PB009 |
| Lower extremity pain | 0 | 1 | 2 | 3 | 4 | PB009 |
| Pain in a dermatome | 0 | 1 | 2 | 3 | 4 | PB009 |
| Pain in another body part (Buttock, hip, groin, thigh) | 0 | 1 | 2 | 3 | 4 | PB009 |
| Generalised pain localisation (3 of 4 body quadrants) | 0 | 1 | 2 | 3 | 4 | PB009 |
| Exercise tolerance (endurance related activities) | 0 | 1 | 2 | 3 | 4 | PD009 |
| Joint mobility | 0 | 1 | 2 | 3 | 4 | PG001 |
| Joint stability | 0 | 1 | 2 | 3 | 4 | PG002 |
| Muscle power | 0 | 1 | 2 | 3 | 4 | PG003 |
| Muscle tone | 0 | 1 | 2 | 3 | 4 | PG003 |
| Muscle endurance | 0 | 1 | 2 | 3 | 4 | PG003 |
| Motor reflex functions (decreased or increased) | 0 | 1 | 2 | 3 | 4 | PG004 |
| Control of movement (Quality, coordination, balance) | 0 | 1 | 2 | 3 | 4 | PG006 |
| Gait pattern | 0 | 1 | 2 | 3 | 4 | PG007 |
| Sensation of muscle stiffness, tightness, spasm, contraction, | 0 | 1 | 2 | 3 | 4 | PG003 |
| heaviness | | | | | | |
| Mobility of spinal meningies, periferal nerves and surrounding | 0 | 1 | 2 | 3 | 4 | PG000 |
| tissue | | | | | | |
| | | | | | | KVÅ |
| 2. Assess grade of <u>ACTIVITY LIMITATION</u> | None | Lite | Moderate | Severe | Complete | code |
| Perception of non-harmful sensory stimuli (kinesiophobia) | 0 | 1 | 2 | 3 | 4 | PJ001 |
| Carrying out daily routine (ADL) | 0 | 1 | 2 | 3 | 4 | PK003 |
| Handling stress and other psychological demands | 0 | 1 | 2 | 3 | 4 | PK004 |
| Changing and maintaining body position (shifting body weight | 0 | 1 | 2 | 3 | 4 | PM001 |
| away from the spine (increased lever arm) | | | | | | |
| Changing and maintaining body position (bending) | 0 | 1 | 2 | 3 | 4 | PM001 |
| Maintaining a lying position | 0 | 1 | 2 | 3 | 4 | PM001 |
| Maintaining a sitting position | 0 | 1 | 2 | 3 | 4 | PM001 |
| Maintaining a standing position | 0 | 1 | 2 | 3 | 4 | PM001 |
| Maintaining an upright neutral posture | 0 | 1 | 2 | 3 | 4 | PM001 |
| Lyfting and carrying objects | 0 | 1 | 2 | 3 | 4 | PM004 |
| Walkning | 0 | 1 | 2 | 3 | 4 | PM007 |
| Moving around in different ways (crawling/climbing, | 0 | 1 | 2 | 3 | 4 | PM008 |
| running/joging, jumping) | | | | | | |
| Household tasks | 0 | 1 | 2 | 3 | 4 | PP003 |
| Work ability and employment | 0 | 1 | 2 | 3 | 4 | PR002 |
| Recreation and leisure activities | 0 | 1 | 2 | 3 | 4 | PS002 |

### DIAGNOSTIC SUBGROUPING AND ICD-10 CODING

- 3. Matching assessment findings to diagnostic codes Choose a primary assessment finding category:
  - First assessment: Cross X one or more related ICD-10 diagnostic codes in the same row
  - Final assessment: Circle O a new diagnostic codes if relevant.

| Primary assessment category | ICD-10 diagnos |
|---|---|
| LBP with muscular functional impairment | ☐ M54.5 Lumbago |
| LBP with segmental mobility impairment | ☐ M54.5 Lumbago ☐ M99.0 Segmental dysfunction |
| LBP with movement coordination impairment/ segmental instability | ☐ M54.5 Lumbago<br>☐ M99.1K Segmental instability in the lumbar<br>spine |
| LBP with referred lower extremity pain (nociceptive pain proximal of the knee) | <ul> <li> □ M54.5 Lumbago □ M51.2 Other specificed dislocation of intervertebral disc □ M47.9K Spondylosis in the lumbar spine </li> </ul> |
| LBP with radiating pain (neuropathic pain) | ☐ M54.5 Lumbago<br>☐ M54.1 Radiculopathy (femoralis)<br>☐ M54.4 Lumbago with ischias |
| LBP with related cognitive or affective tendensies | ☐ M54.5 Lumbago<br>☐ G96.8 Other specified disorders of the CNS<br>(pain sensitivity) |
| LBP with related generaliserad pain (pain in 3 of 4 body quadrants) | <ul> <li>□ M54.5 Lumbago</li> <li>□ G96.8 Other specified disorders of the CNS</li> <li>(pain sensitivity)</li> <li>□ F45.4 Chronic somatoform pain syndrome</li> </ul> |
| LBP with postural related symptoms | ☐ M54.5 Lumbago<br>☐ M40.3 Flatback syndrome<br>☐ M40.4 Hyperlodosis |
| SI-joint symptoms or Coccygodynia | ☐ M53.3 Sacrococcygeal disorders |
| LBP radiating pain + Medical imaging disc pathology and nerve compression finding | ☐ M51.1K Disc degeneration/disc herniation in the lumbar spine with radiculopathy |
| LBP with radiating pain/neurogenic claudication + Medical imaging verifieried degeneration and nerve compression findings | <ul> <li>□ M48.0K Central spinal stenos in the lumbar spine (bilateral symptoms)</li> <li>□ M99.6 Stenosis of intervertebral foramin (unilateralt symptoms)</li> </ul> |
| Ländryggsbesvär med nedsatt rörelse kontroll i<br>ryggen och/eller segmentell instabilitet + Medicinsk<br>bild verifierad Spondylolys/Spondylolisthes | ☐ M43.0 Spondylolys ☐ M43.1 Spondylolistes |

### **TREATMENT**

### 4. Record at final assessment:

| Has the BetterBack☺ model of care Part 1 bee | - ' ' | ☐ Yes ☐ No |
|---|---|---|
| Has the BetterBack© model of care Part 2 bee | ☐ Yes ☐ No | |
| | Cross X all modes och types of treatments used | |
| Physical exercise | MODE | KVÅ code |
| | ☐ Non-supervised individual training | |
| | ☐ Supervised individual training | QV011 |
| | ☐ Supervised group training | QV012 |
| | TYPE | |
| | ☐ Muscle strengthening training | QG003 |
| | ☐ Range of movement training | QG001 |
| | ☐ Muscle endurance training | QG003 |
| | ☐ Cardiovascular training | QD016 |
| | ☐ Balance training | QB001 |
| | ☐ Postural control training | QG004 |
| | ☐ Coordination training | QG005 |
| | ☐ Pelvic floor training | QF001 |
| | ☐ Postural training | QM005 |
| | ☐ Relaxation training | QG007 |
| | ☐ Physical activity prescription (FaR®) | DV002 |
| | ☐ Other | |
| Behavioural medicine interventions | MODE | |
| | ☐ Individual based intervention | QV011 |
| | ☐ Group based intervention | QV012 |
| | TYPE | |
| | ☐ Information / education on pain | QV007 |
| | □ Cognitive-behavioural therapy | DU011 |
| | □ Mindfulness | DU032 |
| | ☐ Motivational interviewing | DU118 |
| | ☐ Relapse prevention | DU119 |
| | ☐ Supportive conversation | DU007 |
| | □ Other | |
| Manual therapy | TYPE | |
| ivialidal therapy | ☐ Joint mobilisation | DN006 |
| | ☐ Joint mobilisation | DN008 |
| | ☐ Massage | QB007 |
| | ☐ Stretching | DN009 |
| | ☐ Nerve mobiliseration | QG001 |
| | ☐ Trigger point pressure | DN007 |
| | ☐ Traction | QG001 |
| | □ Other | Q0001 |
| Occupational medicine interventions | TYPE | + |
| Occupational medicine interventions | ☐ Workplace training | DV084 |
| | ☐ Training of work ability | QR003 |
| | ☐ Work and employment counciling | QR002 |
| | ☐ Information /education on ergonomics | QV010 |
| | Other | QVUIU |
| Physical modalities | TYPE | |
| i nysicai modalities | □ TENS | DA021 |
| | ☐ Cryotherapy | QB011 |
| | ☐ Heat | QB011 |
| | □ Ultrasound | QB011 |
| | ☐ Shockwave therapy | QB011 |
| | ☐ Laser therapy | QB011 |
| | ☐ Short wave diathermy | DV042 |
| | ☐ Interferential therapy | DA021 |
| | □ Orthosis | DN003 |
| | ☐ Taping | DN003 |
| | ☐ Bio-feedback | DV010 |
| | ☐ Acupunkture | DA001 |
| | □ Other | 5,001 |
| 5. Rate overall treatment effect | ☐ Much better | |
| J. Nate Overall treatment effect | Quite much better | |
| | ☐ Unchanged | |
| | ☐ Quite much worse | |
| | ☐ Much worse | |
| | • | |

### 5. Clinical reasoning and process pathway for therapists

A thorough history and adequate physical examination are of great importance in order to target treatment interventions. In addition, it is very important to exclude the few red flag cases that require acute medical or specialist referral for the investigation and treatment of tumors, infections, inflammatory diseases, more severe back pathology and neurological conditions, as well as the strong influence of psychosocial factors which can also cause back pain. StarT Back Tool can be used to support decision making regarding the extent of health care needed and the need for psychosocial focus based on an assessment of risk factors for continued back pain. The physical assessment should include an analysis of functional movements, posture, active movements, passive movements, combined movements and / or static positions, joint accessory movement / provocation tests and neuromuscular function. This is to investigate how the symptoms are related to motion dysfunction.

Based on assessment findings, relevant treatment measures with effect mechanisms directed at functional impairments and activity limitations should be tested. These may include range of movement exercises (active/passive or accessory joint mobilisation or neuromuscular structure mobilisation), motor control exercises, muscle stretching, balance exercises, coordination, muscle strength, muscle endurance, general physical fitness or cardiovascular exercise. For example:

- 1. In the identification of movement directions and positions that reduce or centralize the patient's localised pain, distal pain or radiculopathy, these may be considered as a treatment techniques. This allows the patient to learn strategies to control pain and thus take better responsibility for his or her own situation.
- 2. In the identification of movement restriction due to joint, muscle or nerve related impairment, mobilisation strategies for the relevant structure may be considered to reduce the movement restriction.
- 3. In the identification of segmental instability or trunk motor control impairment in the, exercises with a focus on movement control can be tested aiming to improve muscle function, reduce pain and optimise loading of the trunk during full body movement.
- 4. In the identification of a psychogenic causes of back pain, supervised exercise could be tested to minimize kinesiophobia. This can often be complemented with patient education that can help pain management and enable self-care.
- 5. In the identification of a postural impairment, posture correction and ergonomic interventions can be tested.

Dosage of treatment measures should be individualised and sufficient to achieve the desired effect. Initial targeted treatment should be through individual patient care. As a complement to the initial targeted treatments, the purpose of a general training and patient education is to restore or improve function and activity. The suitability of group-based patient care is assessed in consultation with the patient as general training and patient education is considered relevant to support the patient's self-care.



# **BetterBack** Information on Low Back Pain







### Low Back Pain

Low back pain (LBP) is a common harmless condition that affects almost everyone at some point. Over a one-year period, 4 out of 10 adults experience LBP. It is often characterised by varying degrees of pain and discomfort that may impact on ability to perform activities. An episode of LBP usually improves within 2-6 weeks. Most have a fairly stable pattern of back health for many years, which may sometimes be interrupted by a period of LBP. This is a normal pattern and does not mean that the condition is getting worse over time.

### Degenerative changes in the spine

Something that astonishes many is that there is no direct connection between degenerative changes in the spine and common LBP. This means that changes seen on X-rays, magnetic cameras and computer tomography can show pronounced age related changes or disc herniation in a completely painless person, while someone with LBP may have very little or no changes.

### The structure and function of the lower back and common causes of LBP

The lower back consists of many structures such as bones, joints, discs, stabilising ligaments, nerves, as well as deep and superficial muscles. Pain sensations may potentially be signalled by one or more structures of the lower back. It is often difficult to specify exactly if and which structures signal pain sensations. How we maintain an upright position in different situations is called posture. An optimal posture means that the spine has the best conditions for good mobility with optimal distribution of body weight. Suboptimal posture, suboptimal loading of the back or even too little loading of the back can be possible contributing factors of LBP.

### Experience of back pain

Pain is first experienced when interpreted in the brain. How the pain is interpreted depends on experience, thoughts, feelings and expectations. In some cases, pain may be experienced in the lower back but in the absence of pain signals from structures in the lower back. The pain system may also become hypersensitive and in some cases the pain can persist even though the original cause of the pain has resolved.



Figure 1. Pain is interpreted in the brain. This can be in the presence or absence of signals form lower back structures

© Linköping University 20/03/2017

### Back pain symptoms

In addition to back pain, you may have pain in the buttocks and in one or both legs. You may have difficulty standing, sitting, walking, bending etc. This can lead to frustration, depressed mood and anxiety. Some may be afraid of physical activity and become inactive. All of this can impact negatively on you everyday life.

Tips when you have a particularly troublesome period

Think about what you have read in this brochure, that pain comes in periods but usually calms down. Also think about what relieves the symptoms and what you can do when you have a troublesome period. You may have a favorite exercise or other strategy to manage troublesome periods. Contact your physiotherapist for help if you feel after 2-6 weeks that pain doesn't subside. If you have numbness and tingling in both legs, loss of skin sensation or weak muscles in the legs and feet and especially if you have trouble controlling your bladder and bowel you should seek medical care. If you have LBP after an accident or have been previously treated for cancer or osteoporosis, it is also important to seek medical care. For the vast majority, however, back pain is a harmless and common condition that comes and goes.

### **Back Health**

Good back health is a balance between the back's capacity on one side of the scale and physical / mental stresses on the other side as in the figure below.



Figure 2. Balance between back capacity and stresses

Back pain occurs when imbalance occures between back capacity compared to physical / mental stresses as in the figure below.



Figure 3. Imbalance between back capacity compared to physical / mental stresses

### General advice / self-care

During the acute phase, most people are in need to take it easy and adjust their physical and mental stresses. Today, however, there is extensive research that recommends avoiding bedrest and instead modifying physical activity and successively returning to normal activities as quickly as possible. You can use a pain management scale to find the right level of back physical and mental stresses during everyday activities and also when you work out. This model is based on keeping you within acceptable perceived pain levels during an activity and within 24 hours after activity. This means that activity may increase the pain within acceptable pain levels during or after training, but it should return to initial levels within 24 hours. If you are unsure about the right level of back physical and mental stresses consult your physiotherapist.



Bild 4. During activity, it is preferable that the pain is within safe to acceptable levels and that the pain returns to initial levels within 24 hours

### Treatment for back pain

The goal is to increase your back's capacity and reduce your physical and mental stresses. You can increase your back's capacity by optimising your back posture, muscle stength, muscle endurance, agility, and improving your overall fitness. You can reduce your physical and mental stresses by optimising your back's physical loads, reducing negative emotions through a positive approach and reducing everyday stress and changing your thoughts about your LBP



Figure 5. How to balance the back's capacity and stresses

### The BetterBack<sup>®</sup> model of care

The BetterBack® model of care for LBP focuses on evidence based physiotherapy, patient education and exercise. The main aim is to manage LBP symptoms and enable the patient's self-care ability. You will receive a thorough assessment and individualised care. Depending on your need for extended support in addition to your physiotherapist's initial interventions, pain education seminars and supervised exercise in a group format can be provided for 6 weeks, 2 times / week. The pain education seminars include explanatory models of what pain is, different ways of managing pain, as well as how to balance your back capacity and your physical and mental stresses you are exposed to. It is common for people to become less physically active after a troublesome period of LBP. It is therefore important to get started with some form of general fitness training. You can improve general fitness by walking, Nordic walking, cycling, jogging and swimming. If you experience pain during activity, you can use the pain management scale (see Figure 4). It is important that you feel motivated and can adapt your training to fit into your everyday life. In the BetterBack® model of care program, you can get help on how to get started!



### 7. BetterBack@ Model part 2 – Group education seminar for patients



# Patient information and education in the BetterBack® model of care

1.Information provided in the broschure

- Epidemiology of LBP
- Low back structure and function
- Possible causes of LBP
- The experience of LBP
- Types of LBP symptoms
- Advice on self-care
- Treatment of LBP
- Information provided in the group education:
- What is pain?
- Different ways to manage pain
- Ideal activity level
- Thoughts about pain
- First aid for pain recurrance



# Main points from the information brochure • LBP i common and harmless • LBP cant be seen on x-ray • Pain is interpreted in the brain in the presence or absence of signals form lower back structures • LBP is an imbalance between back capacity compared to physical / mental stresses Your back's capacity















### Pain experience

- Pain can be dampened
- If you understand it's cause
- If it is predictable
- If you know how to handle the pain
- If it is manageable
- If you have a positive attitude
- If you are goal-focused
- Pain can be aggravated
- If you feel uncertain of its cause
- If it is unpredictable
- If you cant control the pain
- If you have a depressed mood
- If you generally feel pressured
- If it is associated with bad experiences



What dampens / aggravates your pain?





























### Tips...

- Adjust activity and load according to your back capacity, not too much not too little
- · Distribute activity throughout the day
- · Be active, take short breaks
- · Think positive thoughts
- Help yourself
- · And ask for help from others





# Increase your capacity – improve general fitness

Help yourself to be physically active to optimising brain and body's wellbeing.

- · Improved memory & concentration
- Better coping with stress
- Improved mood
- Divert negative thoughts
- Contributes to better health, physical and mental















### 8. BetterBack@ Model – Training program for patients

| Training pro | Training program for patients receiving the BetterBack⊕ model of care for LBP | |
|---|---|---|
| Part 1: Posture,<br>muscle control and<br>coordination of basic<br>body movements | Goal: To ensure the patient has satisfactory posture and trunk muscle activation in static positions as well as in conjunction with basic body movement in the sitting, sitting and standing. Implementation*: Exercises and dosages are individually adjusted by the treating therapist. Exercises are performed as home programs and daily training is recommended for optimal results. The therapist assesses when basic competencies in program 1 are achieved before progressing to program 2. | Training range of movement Goal: Restore normal mobility. Implementation: Individualise based on if the patient has movement |
| Part 2: Graded training of muscle strength, coordination and endurance | Goal: To ensure the patient has satisfactory ability to perform more challenging body movements with adequate strength, corrdination and endurance. Implementation*: Exercises and dosages are individually adjusted by the treating therapist. Exercises are performed twice a week for 12 weeks with follow-up conducted by the treating therapist. During the first 6 weeks, patients are offered the opportunity to train in a group supervised by a physiotherapist. The patient will then receive support and feedback regarding the practice of exercises and help to upgrade exercises if necessary. Patient education on self-care and management of back pain is also performed in groups. | restriction. |

<sup>\*</sup>Prerequisite for upgrading the training program is that the patient can satisfactorily perform basic exercises for posture and trunk control in Part 1. Using Part 2 as a basis, the physiotherapist selects and individualises relevant exercises and dosing based on the assessment findings. If support with the training program is required (in addition to a self-mediated home based program), group training supervised by another therapist can implemented. However, the follow-up of the patient is still the responsibility of the therapist who first assessed and initiated the patient's treatment plan. The program is designed with graded levels where difficulty level is increased by successively progressing from stages A through to C. Patients are to perform the exercises as instructed. Training can initially produce some muscle soreness, but this is normal and decreases gradually. Contact your physiotherapist if you have questions or feel unsure.

### Part 1. Posture, muscle control and coordination of basic body movements

### 1a. Basic trunk muscle activation and control in a lying position

### Pelvic control exercise

• Lay on your back with your knees bent. Put your hands under your pelvis. Press your lower back down so it flattens down on the surface you are laying on. Feel how the pelvis tilts backwards and has rolled over your hands. Tip the pelvis forward and feel how the lower back rises again. Remove your hands and repeat the tipping forward and backward with less and less movement. Stop when you come to a normal neutral pelvic position.

### Activating your inner trunk muscles

This exercise focuses on the activation of core muscles in your back, abdomen and pelvis. It is also known as "core activation"

- Lay on your back with your knees bent and put your hands on your waist.
- ① Breathe calmly in and out and make an ssss sound and feel your fingers how the inner muscles between your pelvis bones become activated. This muscle activation should be done slowly and with a minimal force where you feel that the lower part of the stomach is pulled inward-backward-upward.
  - Alternative instructions
    - Draw the lower part of your stomach inwards from the waist of you pants
    - Imagine that you activate your lower stomach muscles just like if you were tightening av belt around you waist
    - Imagine that your holding on to go to the toalet
- Make sure that **you dont**:
  - o Hold your breath, press your lower back down or bend your back forward



# 1b. Basic trunk muscle activation and control in conjunction with body movement in a lying position

### In conjunction with leg movement

Lay on your back with your knees bent. ① Start with "core activation" ② Move your knee on one side out towards the side with and back to the middle with slow controlled movement. Repeat alternately on each side. Maintain a stable positioning of your trunk and pelvis.

Repetitions\_



Perform the same exercise in side lying with movement of one leg. Perform even on the other side thereafter Repetitions

### In conjunction with arm movement

① Start "core activation". ② Bring your arms up över your head, together or alternately, with slow controlled movement. Maintain a stable positioning of your trunk and pelvis.

Repetitions



### 2a. Basic trunk postural control in a sitting position

With neutral posture, loading of the spine is optimally distributed. Feel how the physical loading on your back increases when you sit with hunched posture, and how it relieves when you hold a neutral posture.

### **Training of posture in sitting position:**

- Sit on a chair with your hands under your buttocks.
- On Rotate your pelvis forward over your hands. You should feel like you are arching your back more. Rock your pelvis backward so you return to a neutral back posture. 
  Rotate your pelvis backwards so that you have a hunched posture. Continue to rotate your pelvis backards and forwards a few times



- Stop in a position where you feel you have a even weight distribution over your hands and neutral back posture.
- Your ears, shoulders and hips should create a straight line vertically.

# 2b. Basic trunk muscle activation in a sitting position

Sit on a chair with good posture. ① Train holding a "core activation".

Repititions



# 2c. Basic trunk muscle activation and control in conjunction with body movement in a sitting position

### In conjunction with leg movement

Sit on a chair or training ball. ① Start with "core activation". ② Lift up your knees alternately with slow controlled movement. Maintain a stable positioning of your trunk and pelvis.

Repetitions



### In conjunction with arm movement

① Start "core activation". ② Bring your arms up över your head, together or alternately, with slow controlled movement. Maintain a stable positioning of your trunk and pelvis.

Repetitions\_



# 3a. Basic trunk postural control in a standing position

With neutral posture, loading of the spine is optimally distributed. Feel how the physical loading on your back increases when you sit with hunched posture, and how it relieves when you hold a neutral posture.

### Training of posture in sitting position:

- Stand with your feet hip width apart
- ① Shift your weight forwards and backwards and find a neutral weight distribution over the soles of your feet.
- ② Bend and straighten your knees a few times and find the position where your knees are slightly bent.
- ③ Tilt your pelvis forwards and backwards a few times and the position in the middle where you pelvis has a neutral position.
- Move your head backwards with your chin in.
- S Bring your shoulders up and then relax your shoulders.
- Your ears, shoulders, hips, knees and feet should now be in a straight line.



# **3b.** Basic trunk muscle activation in a standing position

Stand with a neutral posture. ① Train holding a "core activation".

Antal



3c. Basic trunk muscle activation and control in conjunction with body movement in a standing position.

### In conjunction with weight transfering

Stand with a neutral posture. Place you feet wide apart. ① Start "core activation". ② Transfer your weight from one leg to the other alternately. Maintain a stable positioning of your trunk and pelvis. Repetitions



### In conjunction with arm movement

Stand with a neutral posture. ①Start "core activation". ② Bring your arms up över your head, together or alternately, with slow controlled movement. Maintain a stable positioning of your trunk and pelvis. Repetitions



### Part 2: Graded training of muscle strength, coordination and endurance Difficulty level A **Difficulty level C** Difficulty level B 1A) Pelvis lifts in lying position 1B) Pelvis lifts + leg kicks in lying position 1C) Single leg pelvis lift i lying position Lay on your back with your knees bent and arms by Lay on your back with your knees bent and arms by Lay on your back with your knees bent and arms by your side. your side. vour side. ① Start with "core activation". ① Start with "core activation". ① Start with "core activation". ② Lift up your pelvis from the floor. ② Lift up your pelvis from the floor. ② Lift up your pelvis from the floor and at the Repetitions 3 Lift and extend one leg while maintaining a stable same time lift and extend one leg. Lower your foot positioning of your trunk and pelvis. Lower your foot to the floor again and lower the pelvis. Repeat and to the floor again and lower the pelvis. Repeat and change legs every time. change legs every time. Repetitions each side Repetitions\_ each side Tip: Increase resistance by using theraband placed over you pelvis and hold the ends down with your hands. Tip: Increase resistance by using theraband placed Tip: Increase resistance by using theraband placed over you pelvis and hold the ends down with your over you pelvis and hold the ends down with your hands. hands.

### 2A) Knee lifts in lying position

Lay on your back with your knees bent and put your hands on your waist.

- ① Start with "core activation".
- ② Lift one fot slowly up by bending your hip while maintaining a stable positioning of your trunk and pelvis. Slowly bring your fot back to the floor. Repeat and change legs every time.

Repetitions each side



### 2B) Straight leg raises in lying position

Lay on your back with your knees bent and put your hands on your waist.

- ① Start with "core activation".
- ② Extend and lift one leg while maintaining a stable positioning of your trunk and pelvis. Slowly bring your leg back to the floor. Repeat and change legs every time.

Repetitions each side



### 2C) Rotating sit-ups in lying position

Lay on your back with your knees bent.

- ① Start with "core activation".
- ② Place your hands behind your head and bring your opposite knee and elbow together by bending you back forwards. Repeat alternately on each side.

Repetitions each side



### 3A) Hip muscle training in lying position

Lay on your back with your knees bent and arms by your side. Tie a theraband around your knees.

- ① Start with "core activation".
- ② Move your knees slowly away from each other and slowly back again while maintaining a stable positioning of your trunk and pelvis.

Repetitions\_\_\_\_\_



### 3B) Hip muscle training in side lying position

Lay on your side with your knees bent. Tie a theraband around your knees.

- ① Start with "core activation".
- ② Move your top knee slowly away from the other and slowly back down again while maintaining a stable positioning of your trunk and pelvis.

Repetitions each side



### 3C) Hip muscle training in side lying position

Lay on your side with your legs straignt. Tie a theraband around your ankles.

- ① Start with "core activation".
- ② Move your top leg slowly away from the other and slowly back down again while maintaining a stable positioning of your trunk and pelvis.

Repetitions each side



### Alternative

Stand on one leg in a crouched position. Straighten up and move your free leg diagonally backwards just like skating. Repeat alternately on each side.

### 4A) Side plank + arm movement

Lay on your side with support of your lower arm and knee and lift up your pelvis.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while bringing your free arm up over your head.

The exercise can be done with the pelvis still (static) or by moving the pelvis up and down (dynamically). Perform also on the other side.

Repetitions each side



### 4B) Side plank + arm movement

Lay on your side with support of your lower arm and feet and lift up your pelvis.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while bringing your free arm up over your head.

The exercise can be done with the pelvis still (static) or by moving the pelvis up and down (dynamically). Perform also on the other side.

Repetitions\_\_\_\_\_each side



### 4C) Side plank + arm movement

Lay on your side with support of your lower arm and feet and lift up your pelvis.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while bringing your free arm up and rotating your back.

Repetitions each side



Alternative: Stand beside a therband tied to a pole. Pull the theraband diagonally across your body and rotate your back.

Repetitions each side



### 5A) Chair plank

Stand on your knees and support your lower arms on a chair or pilates ball.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while you lift your knees from the floor. Hold \_\_\_\_\_ seconds. Bring your knees back down to the floor.

Repetitions



### 5B) Floor plank

Stand on your knees and support your lower arms on the floor.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while you lift your knees from the floor. Hold \_\_\_\_\_ seconds. Bring your knees back down to the floor.

Repetitions



### 5C) The plank + leg lifts

Stand on your knees and support your lower arms on the floor.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while you lift your knees from the floor holding your legs straight. Lift one foot up from the floor and hold \_\_\_\_\_\_ seconds. Bring your foot back down to the floor.

Repetitions each side



### 6A) 4-point kneeling superman exercise

Position yourself on your hands and knees with your back straight.

- ① Start with "core activation".
- ② Maintain a stable positioning of your trunk and pelvis while you lift up and down one arm alternately. Try instead one leg alternately. When this is easily accomplished, combined these so that you lift an arm and opposite leg up and down simultaneously and alternate sides.

Repetitions each side



### 6B) 4-point kneeling theraband exercise

Positition yourself on your hands and knees with your back straight. Tie a theraband around your fot and hold on to the other end with your hands.

- ① Start with "core activation".
- ② Lift up and straighten your leg. Hold 5 seconds and then bring your leg down again.

Repetitions each side



### 6C) Superman exercise with theraband

Position yourself on your hands and knees with your back straight. Tie a theraband around your fot and hold on to the other end with your opposite hand.

- ① Start with "core activation", Curl your back and bring your opposite knee and elbow together while holding the theraband.
- ②. Slowly straighten your back, arm and opposite leg to stretch out the theraband. Perform the movement with good control of motion.

Repetitions\_\_\_\_\_each side



Alternativ: Try performing the same exercise while standing on one leg.



### 7A) Push-ups against a wall

- ① Start with "core activation"
- ② Perform push-ups against a wall while maintaining straight back posture.

Repetitions\_\_\_\_\_



### 7B) Push-ups against a table

- ① Start with "core activation"
- ② Perform push-ups against a table while maintaining straight back posture.

Repetitions\_\_\_\_\_



### 7C) Push-ups on the floor

- ① Start with "core activation"
- ② Perform push-ups while maintaining straight back posture.

Repetitions\_\_\_\_\_



Alternativ: Try performing the same exercise with your feet on a pilates ball.



### 8A) Standing arm lifts

Hold on to the ends of a theraband and stand on the middle of theraband

- ① Start with "core activation".
- ② Maintain a straight back posture while you lift your arms up over your head against the resistance of a theraband.

Repetitions\_\_\_\_\_



### 8B) Standing rows

Hold on to the ends of a theraband placed around a pole.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform arm rows alternately from side to side.

Repetitions\_\_\_\_\_



### 8C) Standing straight arm lifts

Hold on to the ends of a theraband and stand on the middle of theraband.

- ① Start with "core activation".
- ② Maintain a straight back posture and straight arms while you lift your arms alternately against the resistance of a theraband.

Repetitions each side



Alternative: Try performing straight arm ski rows.



### 9A) Squats

Stand with your back against the wall or with a pilates ball between your back and the wall. Place your feet hip width apart.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform a squat up to about 90 degrees of knee and hip bending.

Repetitions\_\_\_\_\_



### 9B) Squats with your arms över your head

Stand with your back against the wall or with a pilates ball between your back and the wall. Place your feet hip width apart and your hands över your head.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform a squat up to about 90 degrees of knee and hip bending.

Repetitions\_\_\_\_\_



### 9C) Standing high knee lifts

Stand with your back against the wall, place your feet hip width apart and your arms on the wall.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform high knee lifts with alternating legs.

Repetitions each side



### 10A) Tandem stance lunging weight tranfers

Stand with one foot a step length in front of the other foot.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform weight transfer forwards and backwards from foot to foot. Try even with your other foot forward.

Repetitions each side



### 10B) Lunges

Stand with your feet hip width apart and your arms up horizontal to your body.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform forward lunges by taking av step forward with your weight over that leg och then taking a step back again. Alternate which foot you step forward with.

Repetitions each side



# 10C) Lunges with simultaneous upper body movement

Stand with your feet hip width apart and your arms up horizontal to your body.

- ① Start with "core activation".
- ② Maintain a straight back posture while you perform forward lunges by taking av step forward with your weight over that leg och then taking a step back again. Alternate which foot you step forward with. At the same time as you lung, try lifting upp your arms over your head or rotating your upper body from side to side when holding a stick.

Repetitions each side



### Training range of movement

### 1A) Backward bending (elbow support)

Lay on your stomarch and support yourself on your underarms/elbows. Bend your back backwards by pressing up from your underarms/elbows and return to the start position again.

Repetitions



### 1B) Backward bending (bent arms)

Lay on your stomarch and support yourself with your hands. Bend your back backwards by pressing up from your hands but dont straighten your elbows and thereafter return to the start position again.

Repetitions



### 1C) Backward bending (straight arms)

Lay on your stomarch and support yourself with your hands. Bend your back backwards by pressing up from your hands and straightening your elbows and thereafter return to the start position again.

Repetitions\_



# **2A) Foward bending while laying on your back** Lay on your back and bring your knees up to your

stomach, then return to the start position.

Repetitions\_\_\_\_\_



### 2B) Forward bending on hands and knees

Position yourself on your hands and knees with your back straight. Bend your back forward pressing your lower back upwards while bending your hips and knees so that your knees are in contact with your chest. Return to the starting position.

Repetitions



### 2C) Forward bending in sitting or standing

Stand/sit with your back straight. Starting bending forwards nd bringing your hands down towards the floor. Try to even bend your lower back.
Return to your starting position.

Repetitions\_\_\_\_\_



### 3C) Back roation (full range) 3A) Back rotation (lower back) 3B) Back rotation (lower back and thoracic) Lay on your back and bring your knees down towards Lay on your back and bring your knees down towards Lay on your back and bring your left knee down the floor on onside and then over to the other side. the floor on one side while simultaneously reaching towards the floor on your left side while out with your opposite arm upwards and sidewards. simultaneously reaching out with your left arm Repetitions\_ Change sides by bringing your knees over to the upwards and sidewards. Change sides by bringing each side other side and reach out with your opposite arm your knee over to the other side and reach out upwards and sidewards. with your opposite arm upwards and sidewards. Repetitions each side Repetitions each side Stretching of your buttock muscles Stretching of your hip muscles Before and after exercise, stretching exercises help your muscles. Each stretch can be done several times, with <30 second holds. Here are suggestions for stretching. Stretching of your thigh muscles Stretching of the back of your thighs Stetching of the inside of your thighs/groin

### General training - getting in shape

### Training form

Regular physical exercise as a part of everyday life is important for maintaining good health and fitness. For this, we recommend following a training program prescribed by your physiotherapist. Your training can consist of, for example: walks, nordic walking, cycling, jogging, swimming, dancing, gym. Choose which training form is best for you. You can work out alone or with others in a group. The most important thing is that you feel that you take the time for physical activity in your everyday life.

### **Training intensity**

Training intensity can be regulated through a so-called "pacing model". This means that you slowly and gradually increase your training intensity without overloading. You "pace" yourself in a controlled way to reach your goals. You can monitor your level of exertion by using a scale of 6-20 where the scale is based on your approximate pulse when you multiply by 10.

### You should preferably training with a level of exertion between 11 (fairly light) and 14 (somewhat hard).

You should start exercising at about 20% less duration than you are capacble of. If you feel that the exercise feels very easy (at level 9 or below), you can increase your exercise duration slightly so that you feel at least a farily light exertion level (level 11).

When you experience your exercise exertion is on average under a "somewhat hard" lavel (below 14), you can increase your exercise by 20% after 2 weeks. If you are on level 15 or more, you can continue with the same training for an additional 2 weeks.

When your training duration lasts 30 minutes, you can increase the load by increasing the intensity to 15/16 (Hard - you can not speak on at this intensity) in 10 minute intervals. Then you can increase the number of minutes on this intensity (15/16) every second week.

If you have a bad day, you should work out half of what you planned. In this way you can increase your exercise gradually, without risking doing too much.

### Training Contract:

Training Contract:

I will perform ...... as my training form

I will train 3 times/week

I will begin with ..... minutes

I will increase my training intensity with 20 % every second week until reach my goal capacity.

### Rating of Perceived Exertion Borg RPE Scale How you feel when lying in bed or 6 sitting in a chair relaxed. 7 Very, very light Little or no effort. 8 9 Very light 10 11 Fairly light 12 Target range: How you should feel with exercise or activity. 13 Somewhat hard 15 Hard 17 Very hard How you felt with the hardest work you have ever done. 18 19 Very, very hard

Don't work this hard!

## **Training diary**

Name:

20

Maximum exertion

Your physiotherapist will fill in which exercises you should train. You can cross off when you have

# performed the exercises.

| Week | Part 1 | | | | | | | ] | Better!<br>Pa | Back@<br>rt 2 | 9 | | | | R | terBac<br>lange ( | of<br>ent | General training |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | 1 | 2 | 3 | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 1 | 2 | 3 | Borgskalan |
| | Mon | | | | | | | | | | | | | | | | | |
| | Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri | | | | | | | | | | | | | | | | | |
| | Sat | | | | | | | | | | | | | | | | | |
| | Sun | | | | | | | | | | | | | | | | | |
| | Mon | | | | | | | | | | | | | | | | | |
| | Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri | | | | | | | | | | | | | | | | | |
| | Sat | | | | | | | | | | | | | | | | | |
| | Sun | | | | | | | | | | | | | | | | | |
| | Mon | | | | | | | | | | | | | | | | | |
| | Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri<br>Sat | | | | | | | | | | | | | | | | | |
| | Sat<br>Sun | | | | | | | | | | | | | | | | | |
| | Mon | | | | | | | | | | | | | | | | | |
| | Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri | | | ļ | | | | | | | | | | | | | | |
| | Sat<br>Sun | | | | | | | | | | | | | | | | | |
| | Mon | 1 | | | | | | | | | | | | | | | | |
| | Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri | | | | | | | | | | | | | | | | | |
| | Sat<br>Sun | | | | | | | | | | | | | | | | | |
| | Sun<br>Mon | _ | | | | | | | | | | | | | | | | - |
| | Mon<br>Tue | | | | | | | | | | | | | | | | | |
| | Wed | | | | | | | | | | | | | | | | | |
| | Thu | | | | | | | | | | | | | | | | | |
| | Fri | | | | | | | | | | | | | | | | | |
| | Sat | | | | | | | | | | | | | | | | | |
| | Sun | | | | | | | | | | | | | | | | | |

# **Supplementary file 2**

Summary of the workshop to provide training in the use of the BetterBack<sup>©</sup> model of care.

| Schedule | Content | | Brief description | Learning objectives | BCTs used |
|---|---|---|---|---|---|
| Day 1 | Presentation | | Welcome and introduction | <u> </u> | |
| 08:15- | | | | | |
| 08:30 | | | | | |
| Day 1 | Questionnaire | Participating | Participants receive 20 | To generate | |
| 08:30- | | physiotherapists | minutes to complete the | descriptions recorded | |
| 08:50 | | record | questionnaire | by physiotherapists | |
| | | background | | before and after | |
| | | information, | | BetterBack <sup>©</sup> model of | |
| | | PABQ, PCQ, | | care | |
| | | DIBQ | | | |
| Day 1 | Presentation | LBP clinical | Present evidence based | To understand current | - Instruction on |
| 08:50- | | guidelines | guideline | evidence based | how to |
| 09:40 | | | recommendations and the | recommendations for | perform the |
| | | | development process behind the | primary care of LBP and stakeholder | behavior - Credible source |
| | | | recommendations | involvement in their | - Information |
| | | | recommendations | development | about other's |
| | | | | development | approval |
| Day 1 | Presentation | Background to | Outlines the goals for the | To understand aims, | - Credible source |
| 09:40- | | BetterBack© | day, defines and | objectives and | - Social reward |
| 10:00 | | model of care | conceptualizes the | learning outcomes for | - Pros and cons |
| | | | BetterBack <sup>⊕</sup> model of care | the practitioner | - Comparative |
| | | | and communicates need | education | imagining of |
| | | | for the model of care | | future outcomes |
| Day 1 | Swedish fika | Reflection | Informal discussion about | To evaluate the | - Social support |
| 10:00- | | | aims of the BetterBack☺ | practical aims of the | |
| 10:20 | | | model of care compared to | BetterBack <sup>©</sup> model | |
| Day 1 | Demonstration | Use of | current practice Demonstration of how | To understand how to | - Instruction on |
| 10:20- | Demonstration | implementation | evidence based | practically use | how to |
| 11:40 | | tools | recommendations can be | implementation tools | perform the |
| | | | practically applied in the | to assist clinical | behaviour |
| | | | BetterBack <sup>©</sup> model of care | reasoning for | - Demonstration of |
| | | | | matching assessment | behaviour |
| | | | | findings with | - Problem-solving |
| | | | | appropriate diagnosis | - Feedback on |
| | | | | and treatment | behaviour |
| Day 1 | Reflection | Use of | In pairs, participants | To evaluate the | - Behavioural |
| 11:45- | | implementation | discuss reflections upon | practical use of the | practice/rehearsal |
| 12:00 | | tools | how they can practically | BetterBack© model | |
| | | | apply the implementation tools into their clinical | clinical reasoning tools | Framing/reframing |
| | | | practice | | |
| Day 1 | Lunch break | | practice | | |
| 12:00- | | | | | |
| 13:00 | | | | | |
| Day 1 | Task | Use of | Participants are divided | To develop practical | - Behavioural |
| 13:00- | | implementation | into 3 work groups who | skills in the use of the | practice/rehearsal |
| 14:30 | | tools | each transition between | BetterBack⊕ model | - Feedback on |
| | | | 3x30min patient scenario | clinical reasoning tools | behaviour |
| | | | workstations. Participants | | - Social support |
| | | | practice the application of | | |
| | | | the BetterBack© model | | |
| | | | implementation tools using | | |

| | | | therapist-patient role-play. Feedback is provided from the tutor and between peers | | |
|---|---|---|---|---|---|
| Day 1<br>14:30-<br>15:00 | Task | Feedback on<br>work with<br>patient<br>scenarios | Each group discuss and give<br>feedback on their work<br>with the first patient<br>scenario station (10min per<br>group) | To learn how peers used BetterBack <sup>©</sup> model clinical reasoning tools | - Graded task - Verbal persuasion about capability |
| Day 1<br>15:00-<br>15:20 | Swedish fika | Reflection | Informal discussion about<br>the practical use of the<br>BetterBack <sup>®</sup> model of care<br>compared to current<br>practice | To evaluate the practical use of the BetterBack <sup>®</sup> model clinical reasoning tools | - Social support |
| Day 1<br>15:20-<br>15:40 | Summary of the day | Question and<br>answer<br>session and<br>close | Learning outcomes are summarised | | - Feedback on<br>behaviour |
| Day 2<br>08:15-<br>08:30 | Discussion | | Reflections after the first day of the workshop | | |
| Day 2<br>08:30-<br>09:00 | Presentation | | Benefits of using the implementation tools for assessment, diagnosis and intervention | To appreciate how to practically use implementation tools to assist clinical reasoning for aligning assessment, diagnostics and treatment | - Instruction on how to perform the behaviour - Information about social and environmental Consequences - Credible source - Information about other's approval |
| Day 2<br>09:00-<br>09:20 | Demonstration | BetterBack☺<br>model<br>treatment tools | Patient education (brochure) | To understand how to use the implementation tools for LBP patient education | - Instruction on<br>how to<br>perform the<br>behaviour |
| Day 2<br>09:20-<br>10:00 | Demonstration | BetterBack <sup>©</sup><br>model<br>treatment tools | Group education | To understand how to use the implementation tools for LBP patient education | - Instruction on<br>how to<br>perform the<br>behaviour |
| Day 2<br>10:00-<br>10:20 | Swedish fika | Reflection | Informal discussion about which patients group education is relevant | To reflect on the practical use of the BetterBack <sup>©</sup> model | - Social support |
| Day 2<br>10:20-<br>11:00 | Demonstration | BetterBack©<br>model<br>treatment tools | Exercise program | To understand how to use the implementation tools for an exercise program for LBP | - Instruction on<br>how to<br>perform the<br>behaviour |
| Day 2<br>11:00-<br>12:00 | Task | Use of implementation tools | Participants are divided into 3 work groups who each transition between 3x30min patient scenario workstations. Participants practice the application of the BetterBack© model treatment tools using | To develop practical skills in the use of the BetterBack☺ model treatment tools | - Behavioural<br>practice/rehearsal<br>- Feedback on<br>behaviour<br>- Social support |

| | ı | | | Г | |
|---|---|---|---|---|---|
| | | | therapist-patient role-play. | | |
| | | | Feedback is provided from | | |
| | | | the tutor and between | | |
| D 2 | Lale leneal. | | peers | | |
| Day 2<br>12:00- | Lunch break | | | | |
| 13:00 | | | | | |
| | Taali aantini ad | Use of | Doublein cobe and divided | To develop prostical | Dahariarual |
| Day 2<br>13:00- | Task continued | | Participants are divided into 3 work groups who | To develop practical skills in the use of the | - Behavioural |
| 13:30 | | implementation tools | each transition between | BetterBack© model | practice/rehearsal - Feedback on |
| 13:30 | | toois | 3x30min patient scenario | treatment tools | behaviour |
| | | | workstations. Participants | treatment tools | - Social support |
| | | | practice the application of | | - Social Support |
| | | | the BetterBack© model | | |
| | | | treatment tools using | | |
| | | | therapist-patient role-play. | | |
| | | | Feedback is provided from | | |
| | | | the tutor and between | | |
| | | | peers | | |
| Day 2 | Task | Feedback on | Each group discuss and give | To develop practical | - Graded task |
| 13:30- | | work with | feedback on their work | skills in the use of the | - Verbal |
| 14:00 | | patient | with the first patient | BetterBack⊕ model | persuasion about |
| | | scenarios | scenario station (10min per | treatment tools | capability |
| | | | group) | | , , |
| Day 2 | Demonstration | BetterBack <sup>©</sup> | Display of to navigate the | To understand how to | - Instruction on |
| 14:00- | | model of care | BetterBack☺ model of care | use the BetterBack☺ | how to |
| 14:30 | | website | website | model of care website | perform the |
| | | | | | behaviour |
| Day 2 | Task | Potential future | Participants write on post- | To appreciate the | - Comparative |
| 14:30- | | outcomes of | it notes the most important | potential outcomes of | imagining of |
| 15:00 | | the | future outcomes of the | the BetterBack☺ | future outcomes |
| | | BetterBack☺ | BetterBack <sup>©</sup> model of care | model of care | |
| | | model of care | implementation based on: | | |
| | | implementation | <ol> <li>A professional<br/>perspective</li> </ol> | | |
| Day 2 | Presentation | | 2. A patient perspective Clinical champion presents | To reflect on the | - Action planning |
| 15:00- | Tresentation | | an administrative action | practical use of the | - Action planning |
| 15:30 | | | plan (designed earlier in | BetterBack© model of | |
| 13.30 | | | consensus with clinical | care website | |
| | | | colleagues) for the | care website | |
| | | | implementation of the | | |
| | | | BetterBack© model of care | | |
| | | | at their clinic | | |
| Day 2 | Questionnaire | Participating | Participants receive 20 | To generate | |
| 15:30- | | physiotherapists | minutes to complete the | descriptions recorded | |
| 15:50 | | record | questionnaire | by physiotherapists | |
| | | background | | before and after | |
| | | information, | | BetterBack <sup>©</sup> model of | |
| | | PABQ, PCQ, | | care | |
| | | DIBQ | | | |
| Day 2 | Diploma | | Participants completing the | | - Incentive |
| 15:50- | | | workshop receive a CME | | |
| 16:00 | | | diploma | | |